# The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for study 206854: The Clinical Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/ Vilanterol in a Single Inhaler (TRELEGY™ ELLIPTA™) when Compared with Non-ELLIPTA Multiple Inhaler Triple Therapies in COPD Patients within a Usual Care Setting. |
|---|---|---|
| <b>Compound Number</b> | : | GSK2834425 (GW685698+GSK573719+GW642444) |
| <b>Effective Date</b> | : | 30-Oct-2019 |

# **Description:**

- The purpose of this document is to describe the planned analyses and output to be included in the Clinical Study Report (CSR) for study 206854 (INTREPID: INvestigation of TRELEGY Effectiveness: Usual PractIce Design).
- This RAP is intended to describe the effectiveness and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# **RAP Author(s):**

# Author PPD Statistician, Clinical Statistics

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# • RAP Team Review Confirmations (Method: E-mail):

| Reviewer | Date |
|-------------------------------------------------------|-------------|
| Statistics Leader, Clinical Statistics | 16-Oct-2019 |
| PPD | |
| | 14-Oct-2019 |
| Programming Manager, Clinical Programming | |
| RW Clinical Development Director (CIL) | 13-Oct-2019 |
| PPD | |
| | 14-Oct-2019 |
| Clinical Development Physician (MM) | |
| PPD | 14-Oct-2019 |
| RW Clinical Study Manager (OSL) | 11.0002019 |
| PPD | 15-Oct-2019 |
| Principal Clinical Data Manager (DQL) | 13-001-2019 |
| PPD | 15-Oct-2019 |
| Safety Scientist, SERM, Safety and Medical Governance | 13-00:-2019 |
| PPD | 14 Oat 2010 |
| Global Medical Director, COPD, Respiratory | 14-Oct-2019 |
| PPD | 15 Oct 2010 |
| Director, Patient Reported Outcomes, VEO | 15-Oct-2019 |

# • Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature):

| Approver | Date |
|---|---|
| Senior Statistics Director, Clinical Statistics | 29-Oct-2019 |
| Programming Manager, Clinical Programming (Delegated to PPD , Director Clinical Programming, Statistical Programming & Governance) | 30-Oct-2019 |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DDUCTION | | 7 |
| 2. | CLIMAN | | OCOL INFORMATION | 7 |
| ۷. | | Characa to the Drote | and Defined Chatistical Analysis Diag | |
| | 2.1. | Changes to the Proto | col Defined Statistical Analysis Plan | / |
| | 2.2. | Study Objective(s) ar | nd Endpoint(s) | 8 |
| | 2.3. | | | |
| | 2.4. | Statistical Hypothese | s / Statistical Analyses | 11 |
| 3. | PLAN | NED ANALYSES | | 12 |
| | 3.1. | | | |
| | 3.2. | Final Analyses | | 12 |
| 4. | ANAL | YSIS POPULATIONS . | | 12 |
| | 4.1. | Protocol Deviations | | 13 |
| _ | 00110 | NDEDATIONS FOR D | ATA ANALYOFO AND DATA HANDUNO | |
| 5. | | | ATA ANALYSES AND DATA HANDLING | 14 |
| | 5.1. | | ub-group Display Descriptors | |
| | 5.2. | | | |
| | 5.3. | | | |
| | 5.4. | | riates, Other Strata and Subgroups | |
| | J. <del>T</del> . | | n of Subgroups | |
| | 5.5. | | s and Multiplicity | |
| | 5.6. | | for Data Analyses and Data Handling | 10 |
| | 5.0. | | | 16 |
| 6. | eth in | V DODLII ATIONI ANIAI | _YSES | 17 |
| 0. | 6.1. | | Study Population Analyses | |
| | 0.1. | Overview of Planned | Study Population Analyses | 17 |
| 7. | | | ES | |
| | 7.1. | Primary Effectiveness | s Analyses | 18 |
| | | 7.1.1. COPD Asse | essment Test (CAT) Score | 18 |
| | | 7.1.1.1. E | Endpoint / Variables | 18 |
| | | | Summary Measure | |
| | | | Population of Interest | 18 |
| | | 7.1.1.4. | Strategy for Intercurrent (Post-Randomisation) | |
| | | | Events | |
| | | | Statistical Analyses / Methods | 20 |
| | | 7 | 7.1.1.5.1. Statistical Methodology | 20 |
| | 7.0 | Canadam, Effectives | Specification | |
| | 7.2. | | ess Analyses | |
| | | | iratory Volume in 1 Second (FEV <sub>1</sub> ) | |
| | | | Endpoint / Variables | |
| | | | Summary Measure | |
| | | | Population of Interest | 23 |
| | | | Strategy for Intercurrent (Post-Randomisation) Events | 23 |
| | | | Statistical Analyses / Methods | |

| | | | 7.2.1.5.1. | Statistical Methodology | |
|---|---|---|---|---|---|
| | 700 | Taranala El | <b>-</b> \ | Specification | |
| | 7.2.2. | | | | |
| | | 7.2.2.1. | | Variables | |
| | | 7.2.2.2. | , | Measure | |
| | | 7.2.2.3. | | of Interest | 26 |
| | | 7.2.2.4. | Strategy to | r Intercurrent (Post-Randomisation) | 0.0 |
| | | 7 2 2 5 | | Anglyon / Mothada | |
| | | 7.2.2.5. | | Analyses / Methods | 21 |
| | | | 7.2.2.5.1. | Statistical Methodology | 27 |
| | 7.2.3. | Critical Er | rore (CE) | Specification | 27 |
| | 1.2.3. | 7.2.3.1. | Endpoint / | Variables | 27 |
| | | 7.2.3.1. | | Variables | |
| | | 7.2.3.2. | | of Interest | |
| | | 7.2.3.4. | Strategy fo | r Intercurrent (Post-Randomisation) | 20 |
| | | 1.2.5.4. | Evente | | 28 |
| | | 7.2.3.5. | | Analyses / Methods | |
| | | 7.2.0.0. | | Statistical Methodology | 20 |
| | | | 7.2.0.0.1. | Specification | 20 |
| 7.3. | Other F | ffectiveness | s Analyses | | 32 |
| 7.0. | 7.3.1. | Clinically | Important De | eterioration (CID) | 32 |
| | | 7.3.1.1. | | Variables | |
| | | 7.3.1.2. | | Measure | |
| | | 7.3.1.3. | | of Interest | |
| | | 7.3.1.4. | | r Intercurrent (Post-Randomisation) | |
| | | | | | 32 |
| | | 7.3.1.5. | | Analyses / Methods | |
| | | | | Statistical Methodology | |
| | | | | Specification | 34 |
| | 7.3.2. | Clinically | Important De | eterioration (Analyses of | |
| | | Compone | nts) | | 34 |
| | | 7.3.2.1. | | eduction from Baseline in Trough | |
| | | | | weeks | |
| | | | | Endpoint / Variables | |
| | | | 7.3.2.1.2. | Summary Measure | 35 |
| | | | 7.3.2.1.3. | Population of Interest | 35 |
| | | | 7.3.2.1.4. | Strategy for Intercurrent (Post- | |
| | | | | Randomisation) Events | 35 |
| | | | 7.3.2.1.5. | Statistical Analyses / Methods | 36 |
| | | 7.3.2.2. | | ange (Increase) from Baseline in | |
| | | | | e at 24 Weeks | 37 |
| | | | 7.3.2.2.1. | Endpoint / Variables | |
| | | | 7.3.2.2.2. | Summary Measure | |
| | | | 7.3.2.2.3. | Population of Interest | 37 |
| | | | 7.3.2.2.4. | Strategy for Intercurrent (Post- | |
| | | | 7005- | Randomisation) Events | 37 |
| | 700 | A | 7.3.2.2.5. | Statistical Analysis / Methods | |
| | 7.3.3. | | | oderate/Severe Exacerbations | |
| | 7.3.4. | | | /Severe Exacerbation | |
| 7 1 | 7.3.5. | | | Utilisation (HCRU) | |
| 7.4. | EXDIOLS | iory Enectiv | eness Analy | /ses | 41 |

| | | 7.4.1. | Association of Critical Errors with CAT, Moderate/ Severe Exacerbations FEV <sub>1</sub> and FVC | 41 |
|---|---|---|---|---|
| | | 7.4.2. | Patient Study Experience | |
| | | 7.4.3. | Health Related Quality of Life Questionnaire (HRQoL) | 42 |
| 8. | SAFE | TY ANALY | /SES | 43 |
| | 8.1. | | Events Analyses | |
| | 8.2. | Adverse | Events of Special Interest Analyses | 44 |
| | 8.3. | | afety Analyses | |
| 9. | REFE | RENCES. | | 45 |
| 10. | APPE | | | 46 |
| | 10.1. | | x 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | |
| | | | Exclusions from Per Protocol Population | |
| | 10.2. | | x 2: Schedule of Activities | |
| | | 10.2.1. | Protocol Defined Schedule of Events | 47 |
| | 10.3. | Appendix | x 3: Assessment Windows | 5 <mark>4</mark> |
| | 10.4. | | x 4: Study Phases and Treatment Emergent Adverse | EE |
| | | | Chudy Dhagas | |
| | | 10.4.1. | , | |
| | | | 10.4.1.1. Study Phases for Assessments | |
| | | | 10.4.1.2. Study Phases for Concomitant Medication | |
| | | 10.4.2. | 10.4.1.3. Study Phases for COPD Exacerbations Treatment Emergent Flag for Adverse Events/Serious | 50 |
| | | | Adverse Events | 5 <mark>7</mark> |
| | 10.5. | Appendi | x 5: Data Display Standards & Handling Conventions | |
| | | 10.5.1. | Reporting Process | |
| | | 10.5.2. | | |
| | 10.6. | Appendix | x 6: Derived and Transformed Data | |
| | | 10.6.1. | General | 60 |
| | | 10.6.2. | Study Population | 60 |
| | | 10.6.3. | Effectiveness | 6 <mark>5</mark> |
| | | 10.6.4. | Safety | 71 |
| | 10.7. | Appendix | x 7: Reporting Standards for Missing Data | 72 |
| | | | Premature Withdrawals | 72 |
| | | 10.7.2. | | |
| | | | 10.7.2.1. Handling of Missing and Partial Dates | |
| | 10.8. | Appendi | x 8: Abbreviations & Trade Marks | |
| | | 10.8.1. | | |
| | | 10.8.2. | Trademarks | |
| | 10.9. | Appendix | x 9: List of Data Displays | |
| | | 10.9.1. | Data Display Numbering | |
| | | 10.9.2. | Mock Example Shell Referencing | |
| | | 10.9.3. | Deliverables | |
| | | 10.9.4. | Study Population Tables | |
| | | 10.9.5. | Study Population Figures | |
| | | 10.9.6. | Effectiveness Tables | |
| | | 10.9.7. | Effectiveness Figures | |
| | | 10.9.8. | Safety Tables | |
| | | 10.9.9. | ICH Listings | |

# 

CONFIDENTIAL

2019N418769\_00

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report (CSR) for study 206854 for Protocol:

| Revision Chronology: | | |
|----------------------|-------------|-------------|
| 2017N321744_00 | 06-NOV-2017 | Original |
| 2017N321744_01 | 15-FEB-2018 | Amendment 1 |
| 2017N321744_02 | 28-SEP-2018 | Amendment 2 |

Note that in line with the Protocol, this RAP will use the term "Participant" (except Appendix 9: List of Data Displays), while all data displays (Tables, Figures & Listings) produced as part of the planned dry-run and the Statistical Analysis Complete (SAC), will use the term "Subject" which reflects GSK Data Display Standards terminology.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the original protocol (Dated: 06-NOV-2017), protocol amendment 1 (Dated: 15-FEB-2018) and protocol amendment 2 (Dated 28-SEP-2018) are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Other Endpoint: Proportion of responders who experience CID. (Section 2.2) | Other Endpoint: Proportion of participants who experience CID. | The CID is a negative outcome and so the use of word "responder" may be misleading. Wording has been updated in the RAP to avoid misinterpretation. |
| Exploratory Endpoint: Numerical correlation of CE with CAT, moderate/severe exacerbations and FEV <sub>1</sub> (Section 2.2) | Exploratory Endpoint: Association of CE with CAT score, moderate/ severe exacerbations, FEV <sub>1</sub> and FVC | No formal statistical analysis was planned for this exploratory endpoint. Association between the endpoints will be investigated through graphical representation of the data and data summarisation (frequency tables as defined in Section 7.4.1) |
| Analysis Populations - FEV1: All members of the ITT population for whom an FEV <sub>1</sub> assessment was planned. | Analysis Populations - FEV <sub>1</sub> : All members of the ITT population for whom a spirometry assessment was performed at any of Visit 1 or | Change of population definition to be consistent with the information collected in the study eCRF. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | Visit 2. Note: If at least a single record exists in the electronic spirometry data provided for a participant then this constitutes evidence that spirometry measurements were taken (or attempted to be taken). The FEV <sub>1</sub> value may still be missing. | |
| Analysis Populations - CE: All members of the ITT population for whom a critical error assessment was planned. Note that participants within selected centres performing inhaler assessments who are not on an inhaler for which an error checklist is available will not be included in this population. | Analysis Populations - CE: All members of the ITT population for whom a critical error assessment was performed at Visit 2. Note: Participants within selected centres performing inhaler assessments who are not on an inhaler for which an error checklist is available will not be included in this population. Also, participants who are on more than one device must perform an assessment for all devices to be included in the population. | Change of population definition to be consistent with the information collected in the study eCRF. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the effectiveness of | Proportion of responders based on the COPD Assessment |
| TRELEGY ELLIPTA with non-ELLIPTA | Test (CAT) at week 24. Response defined as change from |
| MITT for the impact of COPD on wellbeing | baseline of CAT score ≥2 at 24 weeks |
| and daily life after 24 weeks' treatment | |
| Secondary Objectives | Secondary Endpoints |
| To compare the effectiveness of | Change from baseline in FEV <sub>1</sub> at 24 weeks (in a subset of |
| TRELEGY ELLIPTA with non-ELLIPTA | participants) |
| MITT on lung function after 24 weeks' | |
| treatment | |
| To compare critical errors (CE) made by | Percentage of participants making at least 1 critical error in |
| study participants using the ELLIPTA | inhalation technique at 24 weeks (in a subset of participants) |
| inhaler with participants using selected | |
| non-ELLIPTA MITT after 24 weeks' | |
| treatment | |
| Other Objectives | Other Endpoints |
| To compare TRELEGY ELLIPTA with | Proportion of participants who experience CID. CID is a |
| inhaled non-ELLIPTA MITT for a clinically | composite outcome defined as any one of the following |

| Objectives | Endpoints |
|---|---|
| important deterioration (CID) | <ul> <li>events:</li> <li>100 mL reduction from baseline in FEV<sub>1</sub> at 24 weeks</li> <li>An exacerbation (requiring treatment with antibiotics and/or systemic steroids or hospitalisation)</li> <li>2 units change (increase) from baseline in CAT score at 24 weeks</li> </ul> |
| To quantify the incidence, rate and time to first moderate/severe COPD exacerbation for study participants on TRELEGY ELLIPTA compared with participants on non-ELLIPTA MITT | <ul> <li>Annualised rate of moderate/severe exacerbations (defined as: requiring treatment with antibiotics and/or systemic steroids or hospitalisation).</li> <li>Time to first moderate /severe exacerbation (defined as: requiring treatment with one or more of the following: antibiotics, systemic steroids, hospitalisation)</li> </ul> |
| To compare the effectiveness of TRELEGY ELLIPTA with non-ELLIPTA MITT for COPD-related Healthcare Resource Utilisation (HCRU) | <ul> <li>The frequency of COPD related HCRU including:</li> <li>Primary healthcare contacts.</li> <li>COPD related medication.</li> <li>Hospital admissions, outpatient appointments and A&amp;E attendances.</li> <li>Exploratory: frequency of HCRU assessed using electronic health records.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To assess the data for correlation between critical errors and clinical outcomes | Association of CE with CAT score, moderate/ severe exacerbations FEV <sub>1</sub> and FVC |
| To describe the participant study experience | Participant Treatment and Study Satisfaction Questionnaire at 24 weeks/EW Visit. |
| To describe the change from baseline in patient Health Related Quality of Life | Health Related Quality of Life Questionnaire |
| Safety Objectives | Safety Endpoints |
| To compare safety for study participants using the ELLIPTA inhaler with participants using non-ELLIPTA MITT after 24 weeks' treatment | <ul> <li>All serious adverse events</li> <li>Study treatment related adverse events</li> <li>Adverse events that lead to withdrawal from study treatment</li> </ul> |

# 2.3. Study Design



| Overview of St | udy Design and Key Features |
|---|---|
| Treatment | A participant will be assigned a subject number at the time the informed consent is signed |
| Assignment | in accordance with the randomisation schedule. Once a subject number is assigned to a participant it cannot be reassigned to any other participant in the study. The randomisation schedule will be generated using RANDALL NG and all participants will be centrally randomised using an Interactive Web Response System (IWRS), RAMOS NG. |
| | Randomisation (1:1) will be stratified by the " <i>Prior Treatment Therapy</i> " (treatment the participants receive prior to screening; ICS/LABA or LAMA/LABA or ICS/LAMA/LABA) with dynamic blocking allocation by Country. |
| Interim<br>Analysis | No interim analysis is planned. |

# 2.4. Statistical Hypotheses / Statistical Analyses

The primary objective of this study is to evaluate the effectiveness of TRELEGY ELLIPTA versus non-ELLIPTA MITT in COPD patients in a pragmatic setting over 24 weeks. The study will provide evidence to support HCP and payer discussions that TRELEGY ELLIPTA is more effective on CAT improvement than non-ELLIPTA MITT in a patient population representative of everyday clinical practice.

The primary effectiveness outcome is the proportion of CAT responders at week 24 (Visit 2) and the primary treatment comparison is TRELEGY ELLIPTA versus non-ELLIPTA MITT for all participants.

In addition, other exploratory treatment comparisons of TRELEGY ELLIPTA with non-ELLIPTA MITT will be performed for the prior treatment stratification levels of ICS/LABA/LAMA, ICS/LABA and LABA/LAMA separately for the primary outcome only.

The null hypothesis is that there is no difference in the proportion of CAT responders at week 24 between TRELEGY ELLIPTA and non-ELLIPTA MITT:

$$H0: T1 - T2 = 0$$

The alternative hypothesis is that there is a difference between treatment groups:

H1: 
$$T1 - T2 \neq 0$$

where T1 and T2 are, the treatment means for TRELEGY ELLIPTA and non-ELLIPTA MITT respectively.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

There are no interim analyses planned.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.
- 5. Database freeze (DBF) has been declared by Data Management.

This is an effectiveness study that collects data differently to a traditional clinical trial and also allows participants' Investigational Product (IP) to be modified during the study. The trial design (open label) and the ways the study medication data are recorded in the datasets means that steps must be taken to ensure that Statistics and Programming (S&P) remain blinded to study investigator prescribing of study medication until the S&P unblinding (i.e., review of unblinded datasets) takes place at DBR. Formal unblinding via RandALL will occur immediately prior to DBF, per standard practice. Details on the blinding strategy are included in the Blinding Strategy Charter.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses |
|---|---|---|
| | | Evaluated |
| All Subjects | All participants for whom a record exists in the study database, | Study Population |
| Enrolled (ASE) | including screen failures. | |
| Intent-to-Treat | All randomised participants, excluding those who were randomised in | Study Population |
| (ITT) | error. A participant who is recorded as a screen failure and also | Primary, |
| | randomised will be considered to be randomised in error. Any other | Exploratory and |
| | participant who receives a randomisation number will be considered to | Other |
| | have been randomised. Displays will be based on the treatment to | Effectiveness |
| | which the participant was randomised unless otherwise stated. | Safety |
| FEV1 | All members of the ITT population for whom a spirometry assessment | Secondary |
| | was performed at any of Visit 1 or Visit 2. | Effectiveness |
| | Note: If at least a single record exists in the electronic spirometry data | |
| | provided for a participant then this constitutes evidence that spirometry | |
| | measurements were taken (or attempted to be taken). The FEV <sub>1</sub> value | |

| Population | Definition / Criteria | Analyses |
|---|---|---|
| | | Evaluated |
| | may still be missing. | |
| CE | All members of the ITT population for whom a critical error assessment was performed at Visit 2. | Secondary<br>Effectiveness |
| | Note: Participants within selected centres performing inhaler assessments who are not on an inhaler for which an error checklist is available will not be included in this population. Also, participants who are on more than one device must perform an assessment for all devices to be included in the population. | |
| Refer to Appendi | x 9: List of Data Displays which details the population used for each display. | |

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP)

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the Electronic Case Report Form (eCRF).

A listing of any treatment misallocations will be produced for the ITT population.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| 1 | Ellipta FF/UMEC/VI 100mcg/62.5mcg/25mcg<br>QD | FF/UMEC/VI 100/62.5/25 | 1 |
| 2 | Non-Ellipta Multiple Inhaler Triple Therapy (MITT) Usual Care | Non-Ellipta MITT | 2 |
| Treatm | Treatment comparisons will be displayed as follows using the descriptors as specified: | | |
| • FF | FF/UMEC/VI 100/62.5/25 vs Non-Ellipta MITT | | |

# 5.2. Baseline Definitions

For all endpoints, the baseline value will be the value recorded at Visit 1 (Screening & Randomisation).

For the primary endpoint, baseline COPD Assessment Test (CAT) score will be the CAT score recorded at the CAT assessment at Visit 1. Note that for cases where a CAT assessment was not performed at Visit 1 as per Protocol and a historical CAT score was recorded in the eCRF by the Investigator instead, if the date of the historical CAT assessment was more than 14 days prior to Visit 1, then the baseline CAT score data will be considered as missing for the participant and will not be included in the analyses of the primary endpoint.

For the secondary endpoints of  $FEV_1$  and Trough  $FEV_1$ , baseline  $FEV_1$  and baseline Trough  $FEV_1$  will be the pre-bronchodilator  $FEV_1$  and pre-bronchodilator Trough  $FEV_1$  value recorded from the spirometry performed at Visit 1, respectively.

If multiple pre-bronchodilator  $FEV_1$  or Trough  $FEV_1$  records exist for a participant at Visit 1, the latest record that is on or prior to the randomised treatment start date will be considered as baseline (see Section 10.6.3).

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by country and investigative site, unless otherwise specified.

# 5.4. Examination of Covariates, Other Strata and Subgroups

The list of covariates and other strata to be used in statistical analyses is as described in table below, unless otherwise specified in Section 7.

| Category | Details |
|---|---|
| Strata | The study randomisation will be stratified based on the treatment the participants receive prior to screening: ICS/LABA, LABA/LAMA or ICS/LAMA/LABA |
| Covariates | Primary endpoint of CAT score: Baseline CAT score: Number of exacerbations in the prior year (categorical, see Section 10.6.2) Prior medication use strata (actual strata, see Section 10.6.2) Country: Secondary endpoint of FEV1: Baseline FEV1 score Prior medication use strata (actual strata, see Section 10.6.2) Country Timing of Spirometry (see Section 7.2.1.5.1) Secondary endpoint of Trough FEV1: Baseline Trough FEV1 score Prior medication use strata (actual strata, see Section 10.6.2) Country Secondary endpoint of Critical Errors: Country Secondary endpoint of Critical Errors: Country Prior medication use strata (actual strata, see Section 10.6.2) Other endpoint of proportion of participants who experience a CID: Country Prior medication use strata (actual strata, see Section 10.6.2) Baseline Trough FEV1 Baseline CAT score Number of exacerbations in the prior year (categorical, see Section 10.6.2) Consideration will be given around other exploratory covariates for the study endpoints in a supplementary RAP. |

# **5.4.1.** Examination of Subgroups

No subgroups are considered in this RAP. Consideration of subgroups to be used in descriptive summaries and statistical analyses will be given in a supplementary RAP.

# 5.5. Multiple Comparisons and Multiplicity

There is a single primary endpoint and treatment comparison, so no adjustment for multiplicity is required for the primary effectiveness comparison.

With regards to the secondary, other and exploratory endpoints, inference will only be made if the primary analysis achieves significance. Inference for secondary, other or exploratory endpoints will then be made at the 5% significance level. Otherwise results will be for descriptive purposes only.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-to-Treat (ITT) population (as defined in Section 4), unless otherwise specified.

Study population analyses including descriptive statistics of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

In addition, Section 10.6.2 includes details with regards to derivation of data for the study population analyses.

# 7. EFFECTIVENESS ANALYSES

# 7.1. Primary Effectiveness Analyses

# 7.1.1. COPD Assessment Test (CAT) Score

CAT score data are collected at Visit 1 (prior to randomisation) and at Visit 2/ EW visit. If participants are not able to attend the clinic visit at Visit 1, CAT assessment data can be collected at a domiciliary visit instead. If participants are not able to attend the clinic visit at Visit 2, CAT assessment can be performed at a domiciliary visit or at a telephone call.

Visit 1 or Visit 2 CAT score data collected at a domiciliary visit will be used in the statistical analysis and will also be included in data summaries and listings.

Visit 2 CAT score data collected at a telephone call, will not be considered for use in the statistical analyses, unless otherwise stated. This data will not be included in data summaries but will be included in listings.

CAT score data collected during assessments that are considered as EW assessments, will not be considered for use within the statistical analyses, unless otherwise stated. CAT score data collected during EW assessments will be included in data summaries and listings.

#### 7.1.1.1. Endpoint / Variables

The primary endpoint will be the proportion of responders based on CAT at week 24 (Visit 2).

#### 7.1.1.2. Summary Measure

The summary measure used for the treatment comparison will be an Odds Ratio (OR) and a 95% CI

# 7.1.1.3. Population of Interest

The analysis will be based on the Intent-to-Treat (ITT) population (as defined in Section 4), unless otherwise specified.

# 7.1.1.4. Strategy for Intercurrent (Post-Randomisation) Events

The <u>list of intercurrent events/events leading to missing data</u> that may occur during the study and may affect the estimation of the treatment effect are:

- Randomised Treatment Discontinuation: participants may discontinue randomised COPD maintenance therapy and continue in the study without being prescribed another COPD maintenance therapy. This is considered an intercurrent event.
- Randomised Treatment Modification: participants may discontinue randomised COPD maintenance therapy and get prescribed another COPD maintenance therapy during the study. This is considered an intercurrent event.

- **Pulmonary Rehabilitation**: participants may change pulmonary rehabilitation status during the study. E.g., Participant considered to be undergoing pulmonary rehabilitation at Visit 1 but stopped during the study and so no longer on pulmonary rehabilitation at Visit 2. See Section 10.6.3 for definition of pulmonary rehabilitation status at Visit 1 and at Visit 2. This is considered an intercurrent event
- Oxygen Therapy: If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, this is considered as an intercurrent event. If participants start oxygen therapy during the study but they have recorded another oxygen therapy prior to the study start, this is not considered as an intercurrent event.
- Early Withdrawal from Study: participants may prematurely withdraw from the study which results in missing endpoint data.
- Week 24 CAT Score not Available (other reasons than EW): CAT score at week 24 (Visit 2) may not be available for other reasons (not EW).

The strategies for handling these events for this endpoint are described in Table 2.

Table 2 Strategies for handling intercurrent events/events leading to missing data for the primary endpoint of proportion of CAT responders at week 24

| | | Intercurrent | Missin | g Data | | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuatio<br>n | Randomise<br>d Treatment<br>Modificatio<br>n | Pulmonary<br>Rehabilitatio<br>n | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24<br>CAT Score<br>not<br>Available |
| Treatment<br>Policy x<br>Composit<br>e | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | If participants modify their randomised treatment during the study, they will be considered as non-responders for the week 24 CAT score. (Composite) | If participants change pulmonary rehabilitation status during the study, they will be considered as non-responders for the week 24 CAT score. (Composite) | If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, they will be considered as non-responders for the week 24 CAT score. (Composite ) | Missing week 24 CAT score data will be imputed based on the randomised treatment arm characteristics . This assumes MAR. See details in Section 10.7.2. | Missing week 24 CAT score data will be imputed based on the randomised treatment arm characteristics . This assumes MAR. See details in Section 10.7.2. |

This primary estimand for the primary endpoint of week 24 CAT score will assess the randomised treatment effect, handling differently each of the intercurrent events/events leading to missing data described in Table 2 above.

#### 7.1.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.1.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Proportion of responders based on the COPD Assessment Test (CAT) score at week 24 (Visit 2). For definition of CAT responders, see Section 10.6.3.

# **Model Specification**

The primary endpoint of proportion of CAT responders at week 24 will be analysed for the ITT Population using a logistic regression model with treatment as an explanatory variable and baseline CAT score (continuous), number of exacerbations in the prior year (categorical, see Section 10.6.2), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

#### Interaction Testing:

For the primary estimand, interactions between treatment and other factors will be investigated as follows by adding interaction terms to the model defined above.

Separate models will be fitted to investigate the effect of treatment by covariate interactions: (i) with the addition of an interaction term for Treatment by Baseline CAT score, (ii) with addition of interaction term for Treatment by Number of Exacerbations in the Prior Year, (iii) with addition of interaction term for Treatment by Prior Medication Use Strata, (iv) with addition of interaction term for Treatment by Country. **Note:** The logistic regression model described for the primary analysis above will be used, with the addition of each specific interaction term. No multiple imputation will be performed for missing week 24 CAT score data.

The p-value for each interaction test will be presented. If any interaction p-value is less than 0.10 further investigations will be carried out, for example running the analysis by each category of the subgroup. Any outputs from interaction investigation will also be presented.

#### **Model Results Presentation**

The odds ratio, 95% CI and p-value will be presented for the comparison between treatment arms. It will be based on a two-sided hypothesis testing approach of superiority.

#### **Model Checking & Diagnostics**

For the primary estimand, the model assumptions will be assessed by performing a logistic regression analysis using the primary estimand model specified in the *Model Specification* section above. No multiple imputation will be performed for the missing CAT score data at week 24. The Pearson residuals from this

analysis will be plotted.

# Supportive Analyses

Additional supportive estimands will be defined for the primary endpoint of CAT score. The variable/endpoint, the summary measure and the population of interest for the supportive estimands will be as defined in Section 7.1.1.1, Section 7.1.1.2 and Section 7.1.1.3, respectively. The strategies for handling the intercurrent events/events leading to missing data for each of these supportive estimands are as described below:

# **Supportive Estimand I (Treatment Policy x Composite):**

| | | Missir | ng data | | | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuation | Randomised<br>Treatment<br>Modification | Pulmonary<br>Rehabilitation | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24<br>CAT Score<br>not<br>Available |
| Treatment<br>Policy x<br>Composite | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of randomised treatment modification. (Treatment Policy) | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of change of pulmonary rehabilitation status during the study. (Treatment Policy) | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of start oxygen therapy during the study. (Treatment Policy) | If participants prematurely withdraw from study, they will be considered as non- responders for the week 24 CAT score. (Composite) | If week 24 CAT score data are missing for other reasons than EW, participants will be considered as non- responders for the week 24 CAT score. (Composite) |

Supportive Estimand I, will use the actual values of the week 24 CAT score, regardless of whether the intercurrent events described in the table above occurred in the study. A more conservative approach for the missing data will be followed, where participants with missing week 24 CAT score (because of EW or other reasons) will be considered as non-responders (composite strategy).

# Supportive Estimand II (Treatment Policy x Composite):

| | Intercurrent Events | | | | Missing data | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuatio<br>n | Randomise<br>d Treatment<br>Modification | Pulmonary<br>Rehabilitatio<br>n | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24 CAT<br>Score not<br>Available |
| Treatment<br>Policy x<br>Composit<br>e | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. | If participants modify their randomised treatment during the study, they will be considered as non-responders | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of change of pulmonary | Week 24 CAT score data to be used in the analysis regardless of the intercurren t event of start | Missing week 24 CAT score data will be imputed based on the randomised treatment arm characteristics . This assumes | Missing week 24 CAT score data will be imputed based on the randomised treatment arm characteristics . This assumes |

| (Treatment | for the week | rehabilitation | oxygen | MAR. See | MAR. See |
|---|---|---|---|---|---|
| Policy) | 24 CAT | status during | therapy | details in | details in |
| | score. | the study. | during the | Section | Section |
| | (Composite) | (Treatment | study. | 10.7.2. | 10.7.2. |
| | | Policy) | (Treatment | | |
| | | | Policy) | | |

Supportive Estimand II, will use the actual values of the week 24 CAT score, regardless of whether the intercurrent events of randomised treatment discontinuation, change of pulmonary rehabilitation status or start of oxygen therapy have occurred during the study, but a composite strategy will be followed for the intercurrent event of randomised treatment modification. This is to assess the effect of the intercurrent event of randomised treatment modification on the estimate of the treatment effect. The same imputation approach as the one used for the primary estimand (Section 7.1.1.4) will be performed for missing CAT score data at week 24.

# **Supportive Estimand III (Hypothetical):**

| | | Missin | g data | | | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuation | Randomised<br>Treatment<br>Modification | Pulmonary<br>Rehabilitation | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24<br>CAT Score<br>not<br>Available |
| Hypothetical | Ignore actual week 24 CAT score record. Assume is missing at random (MAR) and impute week 24 CAT score as what would have been if participant would not have discontinued from randomised study treatment. | Ignore actual week 24 CAT score. Assume is MAR and impute week 24 CAT score as what would have been if participant would not have modified the randomised treatment. | Ignore actual week 24 CAT score. Assume is MAR and impute week 24 CAT score as what would have been if participant would not have changed pulmonary rehabilitation status. | Ignore actual week 24 CAT score. Assume is MAR and impute week 24 CAT score as what would have been if participant would not have started oxygen therapy. | Missing week 24 CAT score data will be imputed assuming is MAR and impute values as what would have been if participant would not have withdrawn early from study. | Missing week 24 CAT score data will be imputed assuming is MAR and impute week 24 CAT score as what would have been if participant had an available CAT score at week 24. |

Supportive Estimand III, will assess the treatment effect that would have been observed in a hypothetical scenario where no participants experienced the intercurrent events/events leading to missing data described in table above. This method fits a Bayesian normal repeated measures model and then imputes missing week 24 CAT scores assuming that the data is missing at random (i.e. that the participant continues to be treated with their randomised treatment). The imputed and "real"/ available data will be analysed and summarised using Rubin's rules. See details in Section 10.7.2.

# 7.2. Secondary Effectiveness Analyses

# 7.2.1. Forced Expiratory Volume in 1 Second (FEV<sub>1</sub>)

Spirometry data are collected at Visit 1 (pre and post-salbutamol) and at Visit 2/ EW visit (only pre-salbutamol). If participants are not able to attend the scheduled clinic visit at

Visit 1/ Visit 2 to perform the spirometry assessment, the Visit 1/ Visit 2 spirometry assessment can be performed at a domiciliary visit.

Spirometry data collected at a domiciliary visit will be used in the secondary statistical analyses of FEV<sub>1</sub>, unless otherwise stated. This data will also be included in data summaries and listings.

Spirometry data collected during assessments that are considered as EW assessments or have been inadvertently collected during the study and do not qualify as Visit 1/ Visit 2 spirometry, will not be considered for use within the statistical analyses, unless otherwise stated. Spirometry data collected at EW assessments will be included in data summaries and listings. Spirometry data inadvertently collected in the study that do not qualify as Visit 1/ Visit 2 spirometry will not be included in data summaries but will be included in listings.

# 7.2.1.1. Endpoint / Variables

Change from baseline in FEV<sub>1</sub> at 24 weeks.

# 7.2.1.2. Summary Measure

The summary measure will be the adjusted mean treatment differences.

#### 7.2.1.3. Population of Interest

The analysis will be based on the FEV<sub>1</sub> population (as defined in Section 4), unless otherwise specified.

#### 7.2.1.4. Strategy for Intercurrent (Post-Randomisation) Events

The list of <u>intercurrent events/events leading to missing data</u> that may occur during the study and may affect the estimation of the treatment effect are:

- Randomised Treatment Discontinuation: participants may discontinue randomised COPD maintenance therapy and continue in the study without being prescribed another COPD maintenance therapy. This is considered an intercurrent event.
- Randomised Treatment Modification: participants may discontinue randomised COPD maintenance therapy and get prescribed another COPD maintenance therapy during the study. This is considered an intercurrent event.
- **Pulmonary Rehabilitation**: participants may change pulmonary rehabilitation status during the study. E.g., Participant considered to be undergoing pulmonary rehabilitation at Visit 1 but stopped during the study and so no longer on pulmonary rehabilitation at Visit 2. See Section 10.6.3 for definition of pulmonary rehabilitation status at Visit 1 and at Visit 2. This is considered an intercurrent event
- Oxygen Therapy: If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, this is considered as an intercurrent event. If participants start oxygen therapy during the study but

- they have recorded another oxygen therapy prior to the study start, this is not considered as an intercurrent event.
- Early withdrawal from Study: participants may prematurely withdraw from the study which results in missing endpoint data.
- Week 24 FEV<sub>1</sub> Data not Available (other reasons than EW): FEV<sub>1</sub> data at week 24 (Visit 2) may not be available for other reasons (not EW).

The strategies for handling these events for this endpoint are described in Table 3.

Table 3 Strategies for handling intercurrent events/events leading to missing data for the secondary endpoint of change from baseline in FEV<sub>1</sub> at week 24

| | | Missi | ng data | | | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuation | Randomised<br>Treatment<br>Modification | Pulmonary<br>Rehabilitation | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24<br>FEV <sub>1</sub> not<br>Available |
| Treatment<br>Policy | Week 24 FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | Week 24 FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of randomised treatment modification. (Treatment Policy) | Week 24 FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of change of pulmonary rehabilitation status during the study. (Treatment Policy) | Week 24 FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of start of oxygen therapy during the study. (Treatment Policy) | Missing week 24 FEV1 data will be imputed based on the randomised treatment arm. Assumes MAR. See details in Section 10.7.2. | Missing week 24 FEV <sub>1</sub> data will be imputed based on the randomised treatment arm. Assumes MAR. See details in Section 10.7.2. |

This primary estimand for the secondary endpoint of FEV<sub>1</sub> will assess the randomised treatment effect regardless of whether the intercurrent events/events leading to missing data described in Table 3 above have occurred in the study.

#### 7.2.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.2.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Change from baseline in FEV<sub>1</sub> at 24 weeks.

# **Model Specification**

The secondary endpoint of change from baseline in FEV<sub>1</sub> at week 24 will be analysed for the FEV<sub>1</sub> population using an analysis of covariance (ANCOVA) model with treatment as an explanatory variable and baseline FEV<sub>1</sub> (continuous), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

An additional covariate "Timing of Spirometry" (categorical) indicating when the spirometry assessment was performed (i.e., pre/post maintenance COPD therapy) at Visit 1 and Visit 2 will be defined. All possible combinations for timing of spirometry at Visit 1 and Visit 2 will form the levels of the covariate:

| 1 | Visit 1: Pre-COPD maintenance therapy dose – Visit 2: Pre-COPD |
|---|------------------------------------------------------------------|
| | maintenance therapy dose |
| 2 | Visit 1: Pre-COPD maintenance therapy dose – Visit 2: Post-COPD |
| | maintenance therapy dose |
| 3 | Visit 1: Post-COPD maintenance therapy dose – Visit 2: Pre-COPD |
| | maintenance therapy dose |
| 4 | Visit 1: Post-COPD maintenance therapy dose – Visit 2: Post-COPD |
| | maintenance therapy dose |

Interaction between *Treatment* and *Timing of Spirometry* will be checked. If the interaction p-value is less than 0.10 then the estimate of the treatment effect will be based on the model that includes *baseline FEV*<sub>1</sub>, *prior medication use strata*, *country* and the *timing of spirometry* as covariates as well as the interaction term *treatment* by *timing of spirometry*. If the interaction p-value is not less than 0.10 then the estimate of the treatment effect will be based on the model which will only include *baseline FEV*<sub>1</sub>, *prior medication use strata*, *country* and the *timing of spirometry* as covariates.

#### **Model Results Presentation**

Adjusted Least-square (LS) means and LS mean change from baseline values for each treatment group will be presented with their associated standard errors as well as 95% CIs. The estimated treatment difference along with corresponding standard error, 95% CI and p-value will be presented.

#### **Model Checking & Diagnostics**

For the primary estimand, distributional assumptions underlying the model used for analysis will be examined. An ANCOVA analysis will be performed using the primary estimand model specified in the *Model Specification* section above. No multiple imputation will be performed for the missing week 24 FEV<sub>1</sub> data. The normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable, will be produced.

#### 7.2.2. Trough $FEV_1$

Spirometry data will be used in the statistical analyses in the same way as described in Section 7.2.1.

#### 7.2.2.1. Endpoint / Variables

Change from baseline in Trough FEV<sub>1</sub> at 24 weeks. Trough FEV<sub>1</sub> is defined in Section 10.6.3.

# 7.2.2.2. Summary Measure

The summary measure will be the adjusted mean treatment differences.

#### 7.2.2.3. Population of Interest

The analysis will be based on participants included in the FEV<sub>1</sub> population (as defined in Section 4), who also managed to withhold COPD maintenance treatment at both Visit 1 and Visit 2 spirometry assessment (see also Section 10.6.3 for definition of Trough FEV<sub>1</sub>), unless otherwise specified.

# 7.2.2.4. Strategy for Intercurrent (Post-Randomisation) Events

The list of <u>intercurrent events/events leading to missing data</u> that may occur during the study and may affect the estimation of the treatment effect are as described in Section 7.2.1.4.

The strategies for handling these events for this endpoint are described in Table 4.

Table 4 Strategies for handling intercurrent events/events leading to missing data for the secondary endpoint of change from baseline in Trough FEV₁ at week 24

| | | Missing data | | | | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuation | Randomised<br>Treatment<br>Modification | Pulmonary<br>Rehabilitation | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24 FEV <sub>1</sub><br>not Available |
| Treatment<br>Policy | Week 24 Trough FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | Week 24 Trough FEV1 data to be used in the analysis regardless of the intercurrent event of randomised treatment modification. (Treatment Policy) | Week 24 Trough FEV1 data to be used in the analysis regardless of the intercurrent event of change of pulmonary rehabilitation status during the study. (Treatment Policy) | Week 24 Trough FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of start of oxygen therapy during the study. (Treatment Policy) | Missing week 24 Trough FEV <sub>1</sub> data will be imputed based on the randomised treatment arm. Assumes MAR. See details in Section 10.7.2. | Missing week 24 Trough FEV1 data will be imputed based on the randomised treatment arm. Assumes MAR. See details in Section 10.7.2. |

The primary estimand for the secondary endpoint of Trough FEV<sub>1</sub> will assess the randomised treatment effect regardless of whether the intercurrent events/events leading to missing data described in Table 4 have occurred in the study.

# 7.2.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.2.2.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Change from baseline in Trough FEV<sub>1</sub> at 24 weeks.

# **Model Specification**

The secondary endpoint of change from baseline in Trough FEV<sub>1</sub> at week 24 will be analysed for the FEV<sub>1</sub> population using an analysis of covariance (ANCOVA) model with treatment as an explanatory variable and baseline Trough FEV<sub>1</sub> (continuous), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

#### **Model Results Presentation**

Adjusted Least-square (LS) means and LS mean change from baseline values for each treatment group will be presented with their associated standard errors as well as 95% Cls. The estimated treatment difference along with corresponding standard error, 95% Cl and p-value will be presented.

#### **Model Checking & Diagnostics**

For the primary estimand, distributional assumptions underlying the model used for analysis will be examined. An ANCOVA analysis will be performed using the primary estimand model specified in the *Model Specification* section above. No multiple imputation will be performed for the missing week 24 Trough FEV<sub>1</sub> data. The normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable, will be produced.

#### 7.2.3. Critical Errors (CE)

Inhaler error assessment data is collected at a clinic visit at Visit 2/ EW visit. Inhaler error data collected during assessments considered as EW assessments, will not be considered for use within the statistical analyses, unless otherwise stated. Inhaler error assessment data collected during EW assessments will be included in data summaries and listings.

#### 7.2.3.1. Endpoint / Variables

Percentage of participants making at least one critical error in inhalation technique at 24 weeks.

# 7.2.3.2. Summary Measure

The summary measure used for the treatment comparison will be an Odds Ratio (OR) and a 95% CI.

# 7.2.3.3. Population of Interest

The analysis will be based on participants in the Critical Error (CE) population (as defined in Section 4), unless otherwise specified.

#### 7.2.3.4. Strategy for Intercurrent (Post-Randomisation) Events

The following <u>intercurrent events/events leading to missing data</u> are considered for the secondary endpoint of critical errors:

- Randomised Treatment Modification: participants may discontinue randomised COPD maintenance therapy and get prescribed another COPD maintenance therapy during the study. The three following scenarios are considered after the intercurrent event of randomised treatment modification:
  - a) New COPD maintenance therapy uses the same devices as randomised COPD maintenance therapy and error assessments are performed on these new devices.
  - b) New COPD maintenance therapy uses different devices to randomised COPD maintenance therapy, but devices that are assessed in the study (checklists available) and for which error assessments are performed.
  - c) New COPD maintenance therapy uses devices which are not being assessed in this study (no checklists available) and thus no error assessment is available at week 24 (Visit 2).
- Early Withdrawal from Study: participants may prematurely withdraw from the study and so no actual week 24 (Visit 2) inhaler error assessment is performed.
- Week 24 Inhaler Error Assessment Data not Available (other reasons than EW), e.g., participants on multiple inhalers may have missed performing the assessment on the secondary device at week 24 (Visit 2); participant may miss a component of a device assessment and all other question responses indicate correct use.

The strategies for handling these events for this endpoint are described in Table 5.

Table 5 Strategies for handling intercurrent events/events leading to missing data for the secondary endpoint of percentage of participants making at least 1 critical error in inhalation technique at week 24

| | Intercurrent Events | Missing data | |
|---|---|---|---|
| Estimand Randomised Treatment Modification | | Study Withdrawal | Week 24 Inhaler Error<br>Assessment Data not<br>Available |
| Hypothetical | For the purposes of this secondary endpoint analysis any inhaler error assessment data following randomised treatment modification event and falling under scenario a, will be included in the analysis. Any error assessment data following randomised treatment modification and falling under scenario b or c, will be treated as missing (See also Section 10.6.3). | If participant prematurely withdraw from study, no imputation will be performed for the missing actual week 24 inhaler error data. | If week 24 inhaler error data are not available (for other reasons than EW) no imputation will be performed. |

The primary estimand of the secondary endpoint of critical errors will assess the treatment effect that would have been observed in a hypothetical scenario where no participant experienced the intercurrent events/events leading to missing data described in Table 5.

# 7.2.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.3.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Percentage of participants making at least one critical error in inhalation technique at 24 weeks.

# **Model Specification**

The secondary endpoint of percentage of participants making at least one critical error at week 24 will be analysed for the CE population using a logistic regression model with treatment as an explanatory variable. Country (categorical) and prior medication use strata (categorical, see Section 10.6.2) will be included as covariates in the model.

For the non-ELLIPTA MITT arm all devices for which we have error checklists will be considered. Any participant in the non-ELLIPTA MITT arm using a device for which we have no error checklist will not be considered for critical error assessment.

#### **Model Results Presentation**

The odds ratio, 95% CI and p-value will be presented for the comparison between treatment arms. It will be based on a two-sided hypothesis testing approach of superiority.

# Model Checking & Diagnostics

For the primary estimand, the model assumptions will be assessed by plotting the Pearson residuals from this analysis.

# Supportive Analyses

A supportive estimand will be defined for the secondary endpoint of CE. The variable/endpoint, the summary measure and population of interest for the supportive estimands will be as defined in Section 7.2.3.1, Section 7.2.3.2 and Section 7.2.3.3, respectively. The strategies for handling the intercurrent events/events leading to missing data for this supportive estimand are as described below:

#### Supportive Estimand (Treatment Policy)

| | Intercurrent Events | Missing data | |
|---|---|---|---|
| Estimand | Randomised Treatment<br>Modification | Study Withdrawal | Week 24 Inhaler Error<br>Assessment Data not<br>Available |
| Treatment<br>Policy | All available inhaler error assessment data collected at week 24 (Visit 2) will be included in the analysis, regardless of the inhaler device the participants used at the week 24 assessment following the randomised treatment modification event. (Treatment Policy) | If participant prematurely withdrew from study, no imputation will be performed for the missing actual week 24 (Visit 2) inhaler error data. Note: If participant prematurely withdrew from study and an inhaler error assessment was performed at an EW visit, available EW data will be used in the analysis. | If week 24 inhaler error data are not available (for other reasons than EW) no imputation will be performed. |

Supportive Estimand of the secondary endpoint of critical errors will assess the randomised treatment effect regardless of whether the intercurrent events/events leading to missing data described in the table above have occurred in the study.

#### **Exploratory Analyses**

In addition, further exploratory treatment comparisons between the individual inhalers assessed in the study will be performed, if there are at least 100 participants who performed an inhaler error assessment for each of the individual inhalers assessed in the study. The inhaler comparisons to be assessed are:

| Ellipta vs Diskus | Ellipta vs MDI <sup>[1]</sup> |
|-----------------------|-------------------------------|
| Ellipta vs Breezhaler | Ellipta vs Turbuhaler |
| Ellipta vs Handihaler | Ellipta vs Genuair |

- [1] This is for participants whose COPD maintenance therapy is administered via an MDI. Rescue medications administered via an MDI are not included.
- For each of these exploratory comparisons the variable/endpoint and the summary measure will be as defined in Sections 7.2.3.1 and Section 7.2.3.2.
- The population of interest will be participants from the ITT population (as defined in Section 4) with available critical error assessment data on any of the following devices: Ellipta, Breezhaler, Handihaler,

MDI, Turbuhaler, Genuair. <u>Note</u>: Participants whose COPD maintenance treatment is administered via multiple inhalers not all of which have an inhaler error checklist available in the study, but an inhaler error assessment was still performed for any of those that are assessed in the study, then these participants will be included in the population and the available inhaler error data will be use in the analysis (see also Section 10.6.3).

- Intercurrent Events: The inhaler error data at week 24 will be used regardless of the device the
  participants used at the week 24 (Visit 2) assessment following the randomised treatment modification
  event (Treatment Policy).
- Handling Missing Data: Events leading to missing data (e.g., study withdrawal), will be handled as
  described in Section 7.2.3.4, Table 5. This exploratory estimand will assess the device effect on
  participants who remain in the study and provide inhaler error data in any of the devices assessed in the
  study (i.e., devices for which a checklist is available).
- Model Specification: The percentage of participants making at least one critical error at week 24 will be analysed for each inhaler comparison separately, using a logistic regression model with device type as an explanatory variable. Country (categorical) and prior medication use strata (categorical, see Section 10.6.2) will be included as covariates in the model.

# 7.3. Other Effectiveness Analyses

# 7.3.1. Clinically Important Deterioration (CID)

For the endpoint of CID, CAT score data and spirometry data collected at domiciliary visits or at a telephone call (i.e., for CAT at Visit 2) will be used in the statistical analyses as described in Sections 7.1.1 and Section 7.2.1, respectively. CAT score data and spirometry data collected at EW assessments, will be used within the statistical analyses, unless otherwise stated. Spirometry data inadvertently collected in the study that do not qualify as Visit 1/ Visit 2/ EW visit spirometry will not be included in the statistical analyses.

# 7.3.1.1. Endpoint / Variables

Proportion of participants who experience Clinically Important Deterioration (CID). CID is a composite outcome defined in Section 10.6.3.

# 7.3.1.2. Summary Measure

The summary measure used for the treatment comparison will be an Odds Ratio (OR) and a 95% CI.

# 7.3.1.3. Population of Interest

The analysis will be based on the  $FEV_1$  population (as defined in Section 4), unless otherwise specified.

#### 7.3.1.4. Strategy for Intercurrent (Post-Randomisation) Events

The <u>list of intercurrent events/events leading to missing data</u> that may occur during the study and may affect the estimation of the treatment effect are:

- Randomised Treatment Discontinuation: participants may discontinue randomised COPD maintenance therapy and continue in the study without being prescribed another COPD maintenance therapy. This is considered and intercurrent event.
- Randomised Treatment Modification: participants may discontinue randomised COPD maintenance therapy and get prescribed another COPD maintenance therapy during the study. This is considered an intercurrent event.
- **Pulmonary Rehabilitation**: participants may change pulmonary rehabilitation status during the study. E.g., Participant considered to be undergoing pulmonary rehabilitation at Visit 1 but stopped during the study and so no longer on pulmonary rehabilitation at Visit 2. See Section 10.6.3 for definition of pulmonary rehabilitation status at Visit 1 and at Visit 2. This is considered an intercurrent event.
- Oxygen Therapy: If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, this is considered as an

intercurrent event. If participants start oxygen therapy during the study but they have recorded another oxygen therapy prior to the study start, this is not considered as an intercurrent event.

- Early Withdrawal from Study: participants may prematurely withdraw from the study which results in missing endpoint data.
- Week 24 CAT Score Data not Available (other reasons than EW): CAT score at week 24 (Visit 2) may not be available for other reasons (not EW).
- Week 24 FEV<sub>1</sub> Data not Available (other reasons than EW): Trough FEV<sub>1</sub> data at week 24 (Visit 2) may not be available for other reasons (not EW).

The strategies for handling these events for this endpoint are described in Table 6.

Table 6 Strategies for handling intercurrent events/events leading to missing data for the endpoint of proportion of participants who experience CID

| | Intercurrent Events | | | | Missing data | | |
|---|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuatio<br>n | Randomise<br>d<br>Treatment<br>Modificatio<br>n | Pulmonary<br>Rehabilitatio<br>n | Oxygen<br>Therapy | Study<br>Withdraw<br>al | Week 24<br>Trough<br>FEV <sub>1</sub> not<br>Available | Week 24<br>CAT not<br>Available |
| Treatmen<br>t Policy x<br>Composit<br>e | Week 24 Trough FEV <sub>1</sub> data, CAT score data and on-study Exacerbation data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | Week 24 Trough FEV1 data, CAT score data and on-study Exacerbatio n data to be used in the analysis regardless of the intercurrent event of randomised treatment modification . (Treatment Policy) | Trough FEV1 data, CAT score data and on-study Exacerbation data to be used in the analysis regardless of the intercurrent event of change of pulmonary rehabilitation status during the study. (Treatment Policy) | If participant s start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, they will be considered as meeting the criteria for CID. (Composit e) | Missing week 24 Trough FEV1 and CAT score data will be imputed based on the randomise d treatment arm. Assumes MAR. See details in Section 10.7.2. Note: EW data will be included in the analysis. | Missing week 24 Trough FEV <sub>1</sub> data will be imputed based on the randomise d treatment arm. Assumes MAR. See details in Section 10.7.2. | Missing week 24 CAT score data will be imputed based on the randomise d treatment arm. Assumes MAR. See details in Section 10.7.2. |

This primary estimand for the endpoint of proportion of participants who experience CID will assess the randomised treatment effect, handling differently each of the intercurrent events/events leading to missing data described in Table 6 above.

#### 7.3.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.3.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.3.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Proportion of participants who experience a CID. CID is a composite outcome defined in Section 10.6.3.

# **Model Specification**

The endpoint of proportion of participants who experience a CID will be analysed for the  $FEV_1$  population using a logistic regression model with treatment as an explanatory variable and baseline Trough  $FEV_1$  (continuous), baseline CAT score (continuous), number of exacerbations in the prior year (categorical, see Section 10.6.2), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

#### **Model Results Presentation**

The odds ratio, 95% CI and p-value will be presented for the comparison between treatment arms. It will be based on a two-sided hypothesis testing approach of superiority.

#### **Model Checking & Diagnostics**

For the primary estimand, the model assumptions will be assessed by performing a logistic regression analysis using the primary estimand model specified in the *Model Specification* section above. No multiple imputation will be performed for the missing CAT score data or the missing Trough FEV1 data at week 24. The Pearson residuals from this analysis will be plotted.

#### Sensitivity Analyses

A sensitivity analysis will be performed for the estimand defined in Sections 7.3.1.1 to Section 7.3.1.4, using the same model specified for the primary analysis described in the *Model Specification* section above, but excluding the number of exacerbations in the prior year (categorical) from the list of covariates.

<u>Model Specification:</u> The proportion of participants who experience a CID will be analysed for the FEV<sub>1</sub> population using a logistic regression model with treatment as an explanatory variable and baseline Trough FEV<sub>1</sub> (continuous), baseline CAT score (continuous), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

# 7.3.2. Clinically Important Deterioration (Analyses of Components)

Trough FEV<sub>1</sub> data will be used in the analyses as described in Section 7.3.1.

#### 7.3.2.1. 100 mL Reduction from Baseline in Trough FEV<sub>1</sub> at 24 weeks

#### 7.3.2.1.1. Endpoint / Variables

Proportion of participants who experience a 100 mL reduction from baseline in Trough FEV<sub>1</sub> at 24 weeks.

#### 7.3.2.1.2. Summary Measure

The summary measure used for the treatment comparison will be an Odds Ratio (OR) and a 95% CI.

#### 7.3.2.1.3. Population of Interest

The analysis will be based on the  $FEV_1$  population (as defined in Section 4), unless otherwise specified.

# 7.3.2.1.4. Strategy for Intercurrent (Post-Randomisation) Events

The <u>list of intercurrent events/events leading to missing data</u> that may occur during the study and may affect the estimation of the treatment effect are:

- Randomised Treatment Discontinuation: participants may discontinue randomised COPD maintenance therapy and continue in the study without being prescribed another COPD maintenance therapy. This is considered an intercurrent event.
- Randomised Treatment Modification: participants may discontinue randomised COPD maintenance therapy and get prescribed another COPD maintenance therapy during the study. This is considered an intercurrent event.
- **Pulmonary Rehabilitation**: participants may change pulmonary rehabilitation status during the study. E.g., Participant considered to be undergoing pulmonary rehabilitation at Visit 1 but stopped during the study and so no longer on pulmonary rehabilitation at Visit 2. See Section 10.6.3 for definition of pulmonary rehabilitation status at Visit 1 and at Visit 2. This is considered an intercurrent event.
- Oxygen Therapy: If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, this is considered as an intercurrent event. If participants start oxygen therapy during the study but they have recorded another oxygen therapy prior to the study start, this is not considered as an intercurrent event.
- Early Withdrawal from Study: participants may prematurely withdraw from the study which results in missing endpoint data.
- Week 24 Trough FEV<sub>1</sub> Data not Available (other reasons than EW): Trough FEV<sub>1</sub> data at week 24 (Visit 2) may not be available for other reasons (not EW).

The strategies for handling these events for this endpoint are described in Table 7.

Table 7 Strategies for handling intercurrent events/events leading to missing data for the endpoint of proportion of participants who experience a 100mL reduction from baseline in Trough FEV₁ at week 24

| | | Intercurrent | Missing data | | | |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuation | Randomised<br>Treatment<br>Modification | Pulmonary<br>Rehabilitation | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24<br>Trough FEV1<br>not Available |
| Treatment<br>Policy x<br>Composite | Week 24 Trough FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | Week 24 Trough FEV1 data to be used in the analysis regardless of the intercurrent event of randomised treatment modification. (Treatment Policy) | Week 24 Trough FEV <sub>1</sub> data to be used in the analysis regardless of the intercurrent event of change of pulmonary rehabilitation status during the study. (Treatment Policy) | If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, they will be considered as having experienced a 100mL reduction from baseline in Trough FEV1. (Composite) | Missing week 24 Trough FEV <sub>1</sub> data will be imputed based on the randomised treatment arm. Assumes MAR. See details in Section 10.7.2. Note: Trough FEV <sub>1</sub> data collected at EW visits will be included in the analysis. | Missing week 24 Trough FEV <sub>1</sub> data will be imputed based on the randomised treatment arm. Assumes MAR. See details in Section 10.7.2. |

This primary estimand for the endpoint of proportion of participants who experience a 100mL reduction from baseline in Trough FEV<sub>1</sub> at 24 weeks, will assess the randomised treatment effect, handling differently each of the intercurrent events/events leading to missing data described in Table 7 above.

#### 7.3.2.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.3.2.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.
# **Statistical Methodology Specification**

## **Endpoint / Variables**

Proportion of participants who experience a 100 mL reduction from baseline in Trough FEV<sub>1</sub> at 24 weeks.

## **Model Specification**

The endpoint of proportion of participants who experience a 100 mL reduction from baseline in Trough FEV<sub>1</sub> at 24 weeks will be analysed for the FEV<sub>1</sub> population using a logistic regression model with treatment as an explanatory variable and baseline Trough FEV<sub>1</sub> (continuous), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

## **Model Results Presentation**

The odds ratio, 95% CI and p-value will be presented for the comparison between treatment arms. It will be based on a two-sided hypothesis testing approach of superiority.

# **Model Checking & Diagnostics**

For the primary estimand, the model assumptions will be assessed by performing a logistic regression analysis using the primary estimand model specified in the *Model Specification* section above. No multiple imputation will be performed for the missing Trough FEV<sub>1</sub> data at week 24. The Pearson residuals from this analysis will be plotted.

## 7.3.2.2. 2 Units Change (Increase) from Baseline in CAT Score at 24 Weeks

# 7.3.2.2.1. Endpoint / Variables

Proportion of participants who experience a 2-unit change (increase) from baseline in CAT score at 24 weeks.

## 7.3.2.2.2. Summary Measure

The summary measure used for the treatment comparison will be an Odds Ratio (OR) and a 95% CI.

## 7.3.2.2.3. Population of Interest

The analysis will be based on the FEV<sub>1</sub> population (as defined in Section 4), unless otherwise specified.

# 7.3.2.2.4. Strategy for Intercurrent (Post-Randomisation) Events

The <u>list of intercurrent events/events leading to missing data</u> that may occur during the study and may affect the estimation of the treatment effect are:

- Randomised Treatment Discontinuation: participants may discontinue randomised COPD maintenance therapy and continue in the study without being prescribed another COPD maintenance therapy. This is considered an intercurrent event.
- Randomised Treatment Modification: participants may discontinue randomised COPD maintenance therapy and get prescribed another COPD maintenance therapy during the study. This is considered an intercurrent event.

- **Pulmonary Rehabilitation**: participants may change pulmonary rehabilitation status during the study. E.g., Participant considered to be pulmonary rehabilitation at Visit 1 but stopped during the study and so no longer on pulmonary rehabilitation at Visit 2. See Section 10.6.3 for definition of pulmonary rehabilitation status at Visit 1 and at Visit 2. This is considered an intercurrent event.
- Oxygen Therapy: If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, this is considered as an intercurrent event. If participants start oxygen therapy during the study but they have recorded another oxygen therapy prior to the study start, this is not considered as an intercurrent event.
- **Early Withdrawal from Study**: participants may prematurely withdraw from the study which results in missing endpoint data.
- Week 24 CAT Score not Available (other reasons than EW): CAT score at week 24 (Visit 2) may not be available for other reasons (not EW).

The strategies for handling these events for this endpoint are described in Table 8.

Table 8 Strategies for handling intercurrent events/events leading to missing data for the endpoint of proportion of participants who experience a 2-unit change (increase) from baseline in CAT score at week 24

| | | Intercurrent | t Events | | Missin | g data |
|---|---|---|---|---|---|---|
| Estimand | Randomised<br>Treatment<br>Discontinuation | Randomised<br>Treatment<br>Modification | Pulmonary<br>Rehabilitation | Oxygen<br>Therapy | Study<br>Withdrawal | Week 24 CAT<br>not Available |
| Treatment<br>Policy x<br>Composite | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of randomised treatment discontinuation. (Treatment Policy) | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of randomised treatment modification. (Treatment Policy) | Week 24 CAT score data to be used in the analysis regardless of the intercurrent event of change of pulmonary rehabilitation status during the study. (Treatment Policy) | If participants start oxygen therapy during the study and they have not had another oxygen therapy prior to the study start, they will be considered as having experienced a 2 unit increase from baseline in CAT score. (Composite) | Missing week 24 CAT score data will be imputed based on the randomised treatment arm characteristics. This assumes MAR. See details in Section 10.7.2. Note: CAT score data collected at EW visits will be included in the analysis. | Missing week 24 CAT score data will be Imputed based on the randomised treatment arm characteristics. This assumes MAR. See details in Section 10.7.2. |

This primary estimand for the endpoint of proportion of participants who experience a 2-unit change (increase) from baseline in CAT score at 24 weeks, will assess the randomised treatment effect, handling differently each of the intercurrent events/events leading to missing data described in Table 8 above.

# 7.3.2.2.5. Statistical Analysis / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.3.2.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# **Statistical Methodology Specification**

# **Endpoint / Variables**

Proportion of participants who experience a 2-unit change (increase) from baseline in CAT score at 24 weeks.

# **Model Specification**

The endpoint of proportion of participants who experience a 2-unit change (increase) from baseline in CAT score at 24 weeks, will be analysed for the FEV<sub>1</sub> population using a logistic regression model with treatment as an explanatory variable and baseline CAT score (continuous), prior medication use strata (categorical, see Section 10.6.2) and country (categorical) included as covariates.

# **Model Results Presentation**

The odds ratio, 95% CI and p-value will be presented for the comparison between treatment arms. It will be based on a two-sided hypothesis testing approach of superiority.

# Model Checking & Diagnostics

For the primary estimand, the model assumptions will be assessed by performing a logistic regression analysis using the primary estimand model specified in the *Model Specification* section above. No multiple imputation will be performed for the missing CAT score data at week 24. The Pearson residuals from this analysis will be plotted.

#### 7.3.3. Annualised Rate of Moderate/Severe Exacerbations

No formal statistical analysis is planned for the endpoint of the annualised rate of moderate/severe exacerbations and thus no estimands are defined for this endpoint. For derivation of the annualised rate see Section 10.6.3.

Unless otherwise specified, the annualised rate of on-randomised treatment moderate/severe exacerbations as well as the annualised rate of on-study moderate/severe exacerbations will be summarised by the randomised treatment group using descriptive statistics (n, mean, SD, median, min, max), based on the Intent-to-Treat (ITT) population (as defined in Section 4). The COPD exacerbation data will be listed.

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

## 7.3.4. Time to first Moderate/Severe Exacerbation

No formal statistical analysis is planned for the endpoint of the time to first moderate/severe exacerbation and thus no estimands are defined for this endpoint.

Unless otherwise specified, the time to first on-randomised treatment moderate/severe exacerbations as well as the time to first on-study moderate/severe exacerbations will be summarised by the randomised treatment group, based on the Intent-to-Treat (ITT) population (as defined in Section 4), using Kaplan Meir Estimates.

The probability of having a moderate/severe exacerbation with a 95% CI for each treatment group and the median time to event will be presented. Kaplan-Meier curves

will also be presented showing the probability of having an event over time for each randomised treatment group separately plotted on the same figure.

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

# 7.3.5. Healthcare Resource Utilisation (HCRU)

Analyses relating to HCRU outcomes obtained from the Electronic Health Record (EHR) database will be described in a supplementary RAP and reported independently of this RAP.

As part of this RAP, the number of participants who had unscheduled (routine COPD care not included) COPD related healthcare contacts (e.g., deteriorating COPD) and the number of contacts by type (e.g., telephone calls, physician office/practice visits etc) will be summarised by the randomised treatment group.

All available HCRU data collected during the study will be summarised, including data from participants who prematurely withdrew from study.

# 7.4. Exploratory Effectiveness Analyses

# 7.4.1. Association of Critical Errors with CAT, Moderate/ Severe Exacerbations FEV<sub>1</sub> and FVC

No formal statistical analysis is planned for this exploratory endpoint. The association of critical errors with CAT score at week 24 and the association of critical errors with FEV<sub>1</sub> and FVC at week 24 will be graphically presented. In addition, the association of critical errors with change from baseline in CAT score at week 24 and the association of critical errors with change from baseline in FEV<sub>1</sub> and change from baseline in FVC at week 24 will be graphically presented. This will be based on participants in the CE population whose COPD maintenance treatment is administered via inhalers <u>all</u> of which have an inhaler error checklist available in the study.

The association of critical errors with CAT response (i.e., responder vs non-responder) at week 24 will be summarised in a frequency table. In addition, the association of critical errors with on-randomised treatment moderate/severe exacerbations as well as the association of critical errors with on-study moderate/severe exacerbations will be summarised in a frequency table. See also Section 10.6.3.

The CAT score data, spirometry data (i.e., FEV1 and FVC) and critical error data collected at week 24 (Visit 2) will be used for this exploratory endpoint as described in Section 7.1.1, Section 7.2.1 and Section 7.2.3, respectively.

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

# 7.4.2. Patient Study Experience

No formal statistical analysis is planned for the endpoint of Participant Treatment and Study Satisfaction Questionnaire at 24 weeks/ EW Visit.

The participant responses to the Treatment and Study Satisfaction Questionnaire at 24 weeks/ EW Visit will be summarised by the randomised treatment group and listed, based on the Intent-to-Treat (ITT) population (as defined in Section 4), unless otherwise specified. Frequency of the response categories ("Strongly Agree" to "Strongly Disagree") will be presented for each question by randomised treatment group. See also Section 10.6.3.

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

# 7.4.3. Health Related Quality of Life Questionnaire (HRQoL)

No formal statistical analysis is planned for the endpoint of Health Related Quality of Life Questionnaire (HRQoL).

The HRQoL data from each visit (Visit 1 and Visit 2) will be summarised by the randomised treatment group and listed, based on the Intent-to-Treat (ITT) population, unless otherwise specified. For the numerical questions of the questionnaire (Item 2, 3, and 4, see Section 10.6.3) data will be summarised using descriptive statistics (n, mean, SD, median, min, max). For Item 1 of the questionnaire, the frequency of the categories selected at each visit (Visit 1 and Visit 2) will be summarised.

HROoL data collected at an EW visit will also be included in the summaries and listings.

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

# 8. SAFETY ANALYSES

The safety analyses will be based on the Intent-to-Treat (ITT) population (as defined in Section 4), unless otherwise specified.

# 8.1. Adverse Events Analyses

AEs not related to either study treatment or withdrawal from study treatment are not recorded, unless classified as serious adverse events.

Adverse events analyses including the descriptive statistics of Serious Adverse Events (SAEs), study treatment related AEs and AEs that lead to withdrawal from study treatment will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

Serious adverse events (SAEs) associated with study participation or related to any GSK product, will be collected from the point of informed consent until randomisation. All SAEs will be collected from randomisation until completion of the Visit 2/EW Visit, at the time points specified in the Schedule of Activities (SoA) in Section 10.2. Treatment related AEs and AEs leading to study treatment withdrawal, will be collected from randomisation until completion of Visit 2/EW Visit, at the time points specified in the SoA in Section 10.2. All SAEs, and relevant AEs will be summarised and displayed by randomised treatment group. The onset dates of the SAEs/relevant AEs relative to the randomised treatment start and stop dates will be used to determine in which period an AE occurs.

The AE/SAE text recorded in the eCRF will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), and will be reported using the primary System Organ Class (SOC) and Preferred Term (PT). The number of participants with one or more events of any type will be calculated. Results will be displayed in the order of decreasing frequency, both across SOC and within SOC. A SOC will not be included if no SAEs/AEs in that SOC are reported. If the total incidence for any two or more AEs is equal, the events will be presented in alphabetical order.

Adverse events and Serious Adverse Events will also be listed, with SOC, event (PT), treatment group, number of participants with the event, and specific participant numbers. Demographic details (e.g., age, sex and race), as well as details of the individual AEs, will also be included in these listings. Listings will be sorted within participant by the date of onset of the AE.

Note that moderate and severe COPD exacerbation events will be recorded on the Exacerbation page in the participant's eCRF. Because exacerbations are typically associated with the disease under study, an exacerbation will not be reported according to the standard process for expedited reporting of SAEs to GSK unless the event meets any of the criteria defined in Section 9.5.7 of the Protocol.

Details of the SAE/AE summaries and listings are presented in Appendix 9: List of Data Displays.

# 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting. Furthermore, emerging data from on-going studies may highlight additional adverse events of special interest. Therefore, the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.

Serious Adverse Events of Special Interest (SAESI) will be summarised by the randomised treatment arms and by the class of medication taken at the time of the event. SAESI will also be listed. The details of the planned displays are provided in Appendix 9: List of Data Displays.

Table in Section 10.6.4 presents the groups of Serious Adverse Events of Special Interest (SAESI). Groups which are not standardized MedDRA queries (SMQs) comprise a selection of PTs defined by GSK. The complete list, including the PTs that contribute to each of the groups, will be provided by GCSP using the MedDRA version current at the time of reporting. This list will be finalized prior to unblinding the database.

# 8.3. Other Safety Analyses

Any pregnancies reported during the study will be summarised in case narratives. Any pregnancy complication or elective termination of a pregnancy for medical reasons should be recorded as an AE or SAE and included in summaries and listings of AEs/SAEs.

# 9. REFERENCES

GlaxoSmithKline Document Number 2017N321744\_00, Study ID 206854. The Clinical Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in a Single Inhaler (TRELEGYTM ELLIPTATM) when Compared with Non-ELLIPTA Multiple Inhaler Triple Therapies in COPD Patients within a Usual Care Setting. Effective Date 06-NOV-2017.

GlaxoSmithKline Document Number 2017N321744\_01 (Amendment 1), Study ID 206854. The Clinical Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in a Single Inhaler (TRELEGYTM ELLIPTATM) when Compared with Non-ELLIPTA Multiple Inhaler Triple Therapies in COPD Patients within a Usual Care Setting. Effective Date 15-FEB-2018.

GlaxoSmithKline Document Number 2017N321744\_02 (Amendment 2), Study ID 206854. The Clinical Effectiveness of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in a Single Inhaler (TRELEGYTM ELLIPTATM) when Compared with Non-ELLIPTA Multiple Inhaler Triple Therapies in COPD Patients within a Usual Care Setting. Effective Date 28-SEP-2018.

Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2017. Available from: http://goldcopd.org.

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 10.1.1. Exclusions from Per Protocol Population

A per protocol (PP) population is not defined for this study therefore there are no criteria leading to exclusion from a per protocol population. All deviations will be managed during the study according to the PDMP.

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

| PROCEDURE * | | | TREATMENT PE | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| Informed consent form (ICF) | X | | | | | ICF must be signed before any study procedures/assessments |
| Inclusion and exclusion criteria | | X | | | | Recheck clinical status before randomisation and/or 1st prescription for study treatment |
| Demography | | X | | | | |
| Height and weight | | X | | | | |
| Medical history: past and current medical conditions | | X | | | | This includes family history of premature CV disease. |

| PROCEDURE * | | | TREATMENT PE | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| Historical eosinophil count. whole blood count, % eosinophils | X | X | | | | Most recent historical eosinophil measure taken within the <b>previous</b> 36 months prior to patients consenting visit. (Visit 1 or Visit 0 whichever is applicable) • An absolute number of eosinophils and the % of eosinophils out of the total WBC • White Blood Cell count (WBC) |
| Chronic Obstructive<br>Pulmonary Disease<br>(COPD) and<br>Exacerbation history | | X | | | | The number of moderate/ severe exacerbations in the 12 months prior to V1 will be collected. |
| Randomisation | | X | | | | |
| COPD assessment test (CAT) | | X | | X | X | CAT must be completed prior to randomisation and prior to any other study procedures. Participants who have changed or discontinued treatment will remain in the study and complete CAT assessment at the Visit 2/EW Visit. |
| COPD Exacerbation assessment | | | X | X | X | Moderate and severe exacerbations that occur between V1 and V2 will be recorded. |

| PROCEDURE * | | | TREATMENT PE | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| COPD related<br>healthcare resource<br>use assessment | | | X | X | X | Details of primary healthcare contacts, known secondary care contacts and all COPD related medication use that occurs between V1 and V2 will be recorded in the eCRF. |
| Assessment of inhaler errors (subgroup only) | | | | X | X | |
| Spirometry for lung<br>function (subgroup<br>only) | | X | | X | X | Spirometry should be performed before the day's dose of usual care or study medication. The assessment is pre-and post-salbutamol at Visit 1 and pre-salbutamol at Visit 2 /EW Visit. It should be started between approximately 6:00 am and 12:00 pm The most recent use of COPD maintenance inhaler/ study treatment should be noted. |
| Participant treatment & study satisfaction questionnaire | | | | X | X | |

| PROCEDURE * | | | TREATMENT PE | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| Health Related<br>Quality of Life<br>Questionnaire<br>(HRQoL) | | X | | X | X | |
| Review of study<br>treatment related<br>Adverse Events (AE) | | X | X | X | X | Clinical judgment should be used to determine whether there is a relationship between study treatment and each occurrence of each AE/SAE. Study treatment related adverse events must be recorded from V1. Where a causality relationship is determined, this must be recorded as a study treatment related AE. AEs not related to either study treatment or withdrawal from study treatment are not recorded, unless classified as serious adverse events. Refer to Protocol Amendment 2, Appendix 3 for definitions of AEs, SAEs and guidelines on assessment of causality by investigator |

| PROCEDURE * | | | TREATMENT PE | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| Review of Adverse<br>Events (AE) that<br>lead to withdrawal<br>from study treatment | | X | X | X | X | All AEs that lead to withdrawal from study treatment, whether judged related to study treatment or not, should be recorded. The participant should be encouraged to remain in the study for collection of effectiveness and safety data. All AEs that lead to withdrawal from the study whilst the participant is on study treatment, whether judged related to study treatment or not, should be recorded. |

| PROCEDURE * | | | TREATMENT PE | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| SAE review | X | X | X | X | X | SAEs that are related to study participation or to GSK products are collected from the time of consent to randomisation. All other SAEs are recorded from the time of randomisation. Clinical judgment should be used to determine the relationship between study treatment and each occurrence of each AE/SAE. Where a causality relationship is determined, this must be recorded as a study treatment related SAE. Refer to Protocol Amendment 2, Appendix 3 for definitions of AEs, SAEs and guidelines on assessment of causality by investigator. |
| Details of randomised study treatment and any study treatment changes | | X | X | X | X | Reason for change in treatment, details and date of new treatment should be recorded. |

| PROCEDURE * | | | TREATMENT PH | ERIOD | | NOTES |
|---|---|---|---|---|---|---|
| | VISIT 0 Consenting | VISIT 1 Screening & Randomisation | Usual care / contact for COPD related event or serious adverse event | Early<br>Withdrawal<br>(EW) Visit | VISIT 2 | The following sequence of events must be followed 1.ICF, 2. Screening, 3. Randomisation. All three may occur on the same day with no more than 6 weeks between ICF and screening and no more than 6 weeks between screening and randomisation. |
| Study week | | 1 | After week 1 and before Visit 2 | After week 1<br>and before<br>Visit 2 | 24 (±21 days) | EW Visit should only be conducted if the participant discontinues from participating in the study. Participants withdrawing from study treatment but remaining in the study should continue to Visit 2. |
| Details of medicine<br>and therapy taken for<br>respiratory and other<br>selected conditions | | X | X | X | X | |
| | * The timing data. | and number of plans | ned study assessments | s, including asses | sments may | be altered during the study based on newly available |

# 10.3. Appendix 3: Assessment Windows

Clinic visits/phone calls are scheduled to take place as specified in the protocol and the Schedule of Activities table in Appendix 2: Schedule of Activities. All participants should remain in the study and complete the week 24 visit. If this is not possible then an early withdrawal visit should be completed.

If a participant withdraws early from the study and provides early withdrawal assessments (CAT, FEV<sub>1</sub>, Inhaler errors), then consideration is given as to how/if these data are used. This is defined under the estimand framework in the appropriate analysis methodology sections (Section 7).

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 10.4.1. Study Phases

# 10.4.1.1. Study Phases for Assessments

Assessments will be classified according to the time of occurrence relative to the study treatment (i.e., randomised treatment) start/stop date.

| Study Phase | Definition |
|---|---|
| Pre-randomised<br>Treatment | Assessment < Study Treatment Start Date |
| On-randomised<br>Treatment | Study Treatment Start Date ≤ Assessment ≤ Study Treatment Stop Date + 1 |
| Post-randomised<br>Treatment | (Assessment > Study Treatment Stop Date + 1) and (Assessment ≤ Study Conclusion Date) |
| | <u>Note:</u> Participants can prematurely discontinue from the randomised treatment or modify their randomised treatment at any time during the study, at the Investigator's discretion. Any assessment performed after the randomised treatment stop day + 1 and before the study conclusion date will be considered as "Post-randomised Treatment". |
| Post-Study | Assessment > Study Conclusion Date |
| | Note: this post-study data will not be included in any summaries or analyses (but will be listed). |

# 10.4.1.2. Study Phases for Concomitant Medication

Any medication or vaccine for the treatment of a respiratory condition that the participant receives at the time of consent or receives during the study are collected.

Classification of the prior/concomitant medication is described in Table 9.

 Table 9
 Classification of prior/concomitant medication

| | Pre-randomised<br>Treatment | | On-randomised treatment | | Post randomised treatment |
|---|---|---|---|---|---|
| (a)<br>(b)<br>(c)<br>(d)<br>(e)<br>(f)<br>(g)<br>(h)* | x x x x x x x x x x x x x x x x x x x | Treatment Start Date | x<br>x<br>xx | Treatment Stop Date | x<br>x<br>xx |
| (i)*<br>(j)**<br>(k)**<br>(l)<br>(m)*** | ? | Randomised 1 | X | Randomised 7 | x ? |

- x = start/stop date of prior/concomitant medication
- ? = missing start/stop date of prior/concomitant medication

Medications which start/stop on the same day as the randomised treatment start or randomised treatment stop date respectively, will be classed as on-randomised treatment.

Partial dates for concomitant medications (if present) will be imputed as described in Section 10.7.2.1 prior to the classification of the medications as described in Table 9.

Medications that start after the date of study conclusion (i.e., Concomitant Medication Start Date > Study Conclusion Date), will be classified as "Post-Study". This post-study data will not be included in any summaries or analyses but will be listed.

Medications will be grouped based on the Respiratory Medication Class (RMC) (see Section 10.6.2) and sorted in descending order of total incidence for Respiratory Class and in descending order of total incidence for the ingredient within each Respiratory Class. If the total incidence for any two or more ingredients is equal, the ingredients will be presented in alphabetical order.

## 10.4.1.3. Study Phases for COPD Exacerbations

COPD exacerbations will be classified according to the time of occurrence relative to the study treatment (i.e., randomised treatment) start/stop date.

| Study Phase | Definition |
|---|---|
| Pre-randomised<br>Treatment | COPD Exacerbation < Study Treatment Start Date |
| On-randomised<br>Treatment | Study Treatment Start Date ≤ COPD Exacerbation ≤ Study Treatment Stop Date + 1 |
| | Note: If Prior Medication Stop Date = Randomised Treatment Start Date (date overlap) and COPD Exacerbation starts on that day, the COPD exacerbation will be considered as "On-randomised Treatment". |
| Post-randomised<br>Treatment | (COPD Exacerbation > Study Treatment Stop Date + 1) and (COPD Exacerbation ≤ Study Conclusion Date) |
| | Note: Participants can prematurely discontinue from the randomised treatment or modify their randomised treatment at any time during the study, at the Investigator's discretion. Any exacerbation occurring after the randomised treatment stop day + 1 and prior to the study conclusion date will be considered as "Post-randomised Treatment". |
| On-Study | Randomisation Date ≤ COPD Exacerbation ≤ Latest of (Study Conclusion Date or Study Withdrawal Date) |
| Post-Study | COPD Exacerbation > Study Conclusion Date |

<sup>\*</sup> If a medication is stopped on-randomised treatment or post-randomised treatment and no start date is recorded it will be assumed that the medication was ongoing from the pre-randomised treatment phase

<sup>\*\*</sup> If a medication is started pre-randomised treatment or on-randomised treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study

<sup>\*\*\*</sup> If a medication has no start or stop date it will be assumed that the medication was ongoing from the prerandomised treatment phase to the post-randomised treatment phase

| Study Phase | Definition |
|---|---|
| | Note: this post-study data will not be included in any summaries or analyses (but will be |
| | listed). |

# 10.4.2. Treatment Emergent Flag for Adverse Events/Serious Adverse Events

Adverse Events/Serious Adverse Events will be classified according to the time of occurrence relative to the study treatment (i.e., randomised treatment) start/stop date.

| Study Phase | Definition |
|---|---|
| Pre-randomised<br>Treatment | AE/SAE Start Date < Study Treatment Start Date |
| On-randomised<br>Treatment | Study Treatment Start Date ≤ AE/SAE Start Date ≤ Study Treatment Stop Date + 1 |
| | Note: If Prior Medication Stop Date = Randomised Treatment Start Date (date overlap) and AE/SAE starts on that day, the AE/SAE will be considered as "On-randomised Treatment". |
| Post-randomised<br>Treatment | AE/SAE Start Date > Study Treatment Stop Date + 1 |
| | Note: Participants can prematurely discontinue from the randomised treatment or modify their randomised treatment at any time during the study, at the Investigator's discretion. Any AE/ SAEs reported after the randomised treatment stop day +1 and prior to the study conclusion date will be considered as "Post-randomised Treatment". |
| On-Study | Randomisation Date ≤ AE/SAE Start Date ≤ Latest of (Study Conclusion Date or Study Withdrawal Date) |
| Onset Time Since<br>Study Treatment<br>Start Date (days) | <ul> <li>Time since first dose will be derived as followed: <ul> <li>If Study Treatment Start Date or AE/SAE Start Date is missing =&gt; missing</li> </ul> </li> <li>If Study Treatment Start date &gt; AE/SAE Start Date =&gt; AE/SAE Start Date - Study Treatment Start Date</li> <li>If Study Treatment Start Date ≤ AE/SAE Start Date =&gt; AE/SAE Start Date - Study Treatment Start Date + 1</li> </ul> |
| Duration (Days) | AE/SAE Resolution Date – AE/SAE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES'. |

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

# 10.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | : /arenv/arprod/gsk2834425/206854 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK Analysis & Reporting (A&R) dataset standards. | |
| Generation of RTF Files | |
| Rich Text Format (RTF) files will be generated for all Table displays for this reporting effort. | |

# 10.5.2. Reporting Standards

## General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - o 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

**Note:** All data displays (Tables, Figures & Listings) produced as part of the Statistical Analysis Complete (SAC), will use the term "Subject" which reflects GSK Data Display Standards terminology.

#### **Formats**

- All data will be reported according to the treatment the participant was randomised to unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - Actual time will be used for calculation of times to event and Kaplan-Meier plots.
- Reporting for Data Listings:
  - Planned and actual time relative to study start date will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).

# **Unscheduled Visits**

Unscheduled visits will not be included in summary tables and/or figures.

| All unscheduled visits will be included in listings. | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### Study Day

- Calculated as the number of days from Treatment Start Date (i.e., Randomised Treatment Start Date):
  - Reference Date = Missing → Study Day = Missing
  - Reference Date < Treatment Start Date → Study Day = Reference Date Treatment Start Date
  - Reference Data ≥ Treatment Start Date → Study Day = Reference Date (Treatment Start Date)
     + 1

# **Randomised Treatment Start/Stop Date**

 Randomised treatment start date will be defined as the earliest treatment start date and randomised treatment stop date will be defined as the latest treatment stop date as captured in the "Study Treatment" (CONMEDS CR 1) eCRF form.

Missing or partial randomised treatment stop dates will be handled as described in Section 10.7.2.1.

# 10.6.2. Study Population

## Disposition

## **Time to Study Withdrawal/ Treatment Discontinuation**

For Kaplan-Meier plots of study withdrawal over time and discontinuation from study treatment over time, censoring will be performed as follows:

- For study withdrawal, participants are represented from the date of start of the randomised treatment to the date of early withdrawal from the study (or date of death). Participants that completed the study are censored at the earliest of the date of completion and Day 169.
- For discontinuation from study treatment, participants are represented from the date of start of the study randomised treatment to the date of discontinuation from study randomised treatment (or date of death). Participants that complete study randomised treatment are censored at the earliest of their study randomised treatment stop date and Day 169.

# **Demographics**

## Age

- In accordance with GSK policy, only year of birth is collected in the eCRF. In order to estimate participant's age, a complete birthdate will be estimated by using the year recorded in the eCRF and assigning month and day values of '30JUN.'
- Age, in whole years, will be calculated based on the Screening Visit date.
- Birth date will be presented in listings as 'YYYY.'
- Completely missing dates of birth will remain as missing with no imputation applied. Consequently, the age of the participant will not be calculated and will remain missing.

## **Age Categories**

Age categories are based on age at Screening and are defined as:

# **Demographics**

- ≤ 64 years
- 65-74 years
- 75-84 years
- ≥ 85 years

## **Body Mass Index (BMI)**

BMI will be calculated in the eCRF as Weight (kg) / Height (m)2.

### Race

High-level Food and Drug Administration (FDA) race categories and designated Asian subcategories are:

- American Indian or Alaska Native
- Asian
  - Central/South Asian Heritage
  - Japanese Heritage/East Asian Heritage/South East Asian Heritage
  - Mixed Asian Heritage (only required if data exists)
- Black or African American
- Native Hawaiian or other Pacific Islander
- White

These categories and subcategories will be summarised along with all combinations of high-level categories which exist in the data. All five of the high-level race categories and the Asian subcategories must appear on the display even if there are no participants in a particular category, but combinations that do not exist in the data do not need to be represented. Combinations will be represented as the concatenation of the high-level category terms, e.g., "White & Asian". The designated Asian subcategories will not be summarised as combinations with other categories.

In addition, the standard race categories collected per IDSL will be summarized along with categories for mixed race. The categories are:

- American Indian or Alaska Native
- Asian Central/South Asian Heritage
- Asian East Asian Heritage
- Asian Japanese Heritage
- Asian South East Asian Heritage
- Black/African American
- Native Hawaiian or other Pacific Islander
- White Arabic/North African Heritage
- White White/Caucasian/European Heritage
- Mixed Asian Race
- Mixed White Race
- Multiple

"Mixed Asian Race" is only used if more than one Asian category is selected, but no non-Asian races. Similarly, "Mixed White Race" is only used if both of the White categories are selected, and no non-White races. If multiple races of different types are selected, then the overall "Multiple" category is used.

A participant will only be represented in a single category. A participant who selects a combination of races will be counted as "Mixed Asian Race," "Mixed White Race," or "Multiple," but not in each of the constituent terms. Therefore, the counts will add up to the total number of participants with a response.

# **Demographics**

# Age Ranges

For the Summary of Age Ranges, the following ranges will be presented, as per the European Medicines Agency (EMA) clinical trial results disclosure requirements:

- Adults (18-64)
- ≥ 65-84 years
- ≥ 85 years

# **Extent of Exposure and Post-randomised Treatment Study Duration**

• Number of days of exposure to randomised treatment will be calculated based on the formula:

# [ Randomised Treatment Stop Date – Randomised Treatment Start Date ] + 1

Participants who were randomised but did not report a randomised treatment start date will be categorised as having zero days of exposure.

• Duration of post-randomised treatment time spent in the study will be calculated as:

## [ Study Conclusion Date - Randomised Treatment Stop Date ]

• Duration of total time spent in the study will be calculated as:

# [ Study Conclusion Date – Randomisation Date ] + 1

The following exposure categories will also be presented:

 $\geq$  1 day,  $\geq$  4 weeks,  $\geq$  8 weeks,  $\geq$  12 weeks,  $\geq$  16 weeks,  $\geq$  20 weeks,  $\geq$  24 weeks, 23-25 weeks

## **Medical Conditions and Concomitant Medications**

## **COPD Exacerbation History**

- COPD exacerbations occurring in the past 12 months prior to Screening reported on the Exacerbation History eCRF form will be categorized as 0, 1, ≥ 2.
- The number of COPD exacerbations reported in the past 12 months will be summarised according to the categories: 1) moderate COPD exacerbations, 2) severe COPD exacerbations, and 3) moderate/severe COPD exacerbations.

<u>Moderate COPD exacerbations</u>: defined as exacerbations that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization).

<u>Severe COPD exacerbations</u>: defined as exacerbations that required in-patient hospitalization.

<u>Moderate/Severe COPD exacerbations</u>: defined as the total number of moderate and severe COPD exacerbations.

### **COPD Concomitant Medications**

• COPD concomitant medications will be grouped into the following Respiratory Medication Classes (RMC) based on pre-defined code lists derived from Anatomical Therapeutic Chemical (ATC)

## **Medical Conditions and Concomitant Medications**

#### classifications:

- Androgens and estrogens
- o Anti-IgE, Anti-IL5
- Anticholinergic
- Antiinfectives (antibiotics, antiseptics)
- Antimycotics
- Antivirals
- Beta-2 agonists
- Corticosteroid inhaled
- Corticosteroid depot
- Corticosteroid systemic oral parenteral and intra-articular
- Corticosteroid other
- Leukotriene receptor antagonist
- Long-acting anticholinergic
- Long-acting beta-2 agonist Group 2 (once per day)
- Long-acting beta-2 agonist Group 3 (twice per day)
- Mucolytics
- Nedocromil or cromolyn sodium
- o Oxygen
- PDE4 inhibitors
- Short-acting anticholinergic
- Short-acting beta-2 agonist
- Xanthine
- Other COPD medication

# **Actual Prior Medication Use Strata**

The actual prior medication use strata will be defined from the CONMEDS form of the CRF using the COPD maintenance medications taken prior to Randomisation.

## **Historical Eosinophils Data**

Historical Haematology data of White Blood Cell (WBC) and Eosinophils data will be collected at Visit 2. This data will be summarised by the randomised treatment groups (using descriptive statistics) and will be listed. Eosinophils data will also be categorised as described below and summarised by the randomised treatment groups:

- < 0.15 10^9/L</p>
- ≥ 0.15 10^9/L

## **Screening Lung Function**

## Reversibility

A participant's status as reversible to salbutamol is calculated at Screening and is based on the difference (absolute change and % change) between a participant's pre-salbutamol assessment of FEV<sub>1</sub> and their post-salbutamol assessment of FEV<sub>1</sub> and is defined as follows:

- Reversible, if the difference in FEV₁ is ≥ 12% and ≥ 200 mL, or
- Non-reversible, if the difference in FEV₁ is < 200 mL or, the difference is ≥ 200 mL and is < 12 % of the pre-salbutamol FEV₁</li>

If a participant was not able to provide both a pre-salbutamol and post-salbutamol assessment, then the

# **Screening Lung Function**

reversibility status will be missing.

## **GOLD Grade 1-4**

Participants will be classified into Global Initiative on Obstructive Lung Disease (GOLD) Grades 1-4 using the post-salbutamol percent predicted FEV<sub>1</sub> assessment at Screening [GOLD, 2017]:

- GOLD Grade 1 (Mild): percent predicted FEV₁ ≥ 80%
- GOLD Grade 2 (Moderate): 50% ≤ percent predicted FEV<sub>1</sub> < 80%
- GOLD Grade 3 (Severe): 30% ≤ percent predicted FEV<sub>1</sub> < 50%
- GOLD Grade 4 (Very Severe): percent predicted FEV<sub>1</sub> < 30%

If a participant was not able to provide post-salbutamol assessment, then the GOLD Grade will be missing.

## FEV<sub>1</sub>/FVC ratio at Screening

Using the lung function data from the PFT dataset, the following additional calculations will be performed:

• Pre-bronchodilator FEV<sub>1</sub>/FVC ratio will be calculated as:

# [ Pre-bronchodilator FEV<sub>1</sub>/FVC (%) ] / 100

• Post-bronchodilator FEV<sub>1</sub>/FVC ratio will be calculated as:

[ Post-bronchodilator FEV<sub>1</sub> / Post-bronchodilator FVC ]

Pre and post-bronchodilator FEV<sub>1</sub>/FVC ratio at Screening will be summarised.

#### **Cardiovascular Risk Factors**

Participants with at least one of the following current or past medical conditions at Screening will be classed as having a cardiovascular (CV) risk factor.

- Coronary artery disease
- Myocardial infarction
- Arrhythmia
- Congestive heart failure
- Hypertension
- Cerebrovascular accident
- Diabetes mellitus
- Hypercholesterolemia

The number of CV risk factors at Screening  $(0, 1, or \ge 2)$  will be derived.

## 10.6.3. Effectiveness

#### Intercurrent Events

## Pulmonary Rehabilitation Status at Visit 1 and Visit 2

For the Pulmonary Rehabilitation, the following information is collected in the eCRF at Visit 1 and Visit 2:

- V1. Q1: Is the subject currently on a Pulmonary rehabilitation program?
- V1, Q2: Has the subject started a Pulmonary rehabilitation program within the last 8 weeks prior to Visit 1?
- **V1**, **Q3**: Has the subject stopped a Pulmonary rehabilitation program within the last 8 weeks prior to Visit
- **V2**, **Q1**: Is the subject currently on a Pulmonary rehabilitation program?
- **V2**, **Q2**: Has the subject started a Pulmonary rehabilitation program since Visit 1?
- V2, Q3: Has the subject stopped a Pulmonary rehabilitation program since Visit 1?

The Pulmonary Rehabilitation status for a participant at Visit 1 or Visit 2 can be defined as: a) "On Pulmonary Rehabilitation" or b) "Not on Pulmonary Rehabilitation".

- Visit 1: In order for a participant to be considered as "Not on Pulmonary Rehabilitation" at Visit 1, the
  participant should not be currently on a Pulmonary Rehabilitation program at Visit 1 (i.e., <u>All</u> Visit 1
  questions should be answered with a "No").
- Visit 2: In order for a participant to be considered as "Not on Pulmonary Rehabilitation" at Visit 2, the
  participant should not be currently on a Pulmonary Rehabilitation program at Visit 2 (i.e., <u>All</u> Visit 2
  questions should be answered with a "No" <u>and</u> also not considered on Pulmonary Rehabilitation at
  Visit 1).

# **Primary Endpoint**

## **COPD Assessment Test (CAT)**

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are
protected by third party copyright laws and therefore have been excluded.

• For the Effectiveness analysis of CAT score:

If the language of the CAT assessed at week 24 (Visit 2) is different from the language used at baseline (Visit 1), the CAT score at the week 24 (Visit 2) will be set to missing.

With regards to the primary endpoint analyses, a participant will be considered as a responder according to the CAT score if their week 24 (Visit 2) CAT score has decreased at least 2 units from the baseline CAT score. A participant will be considered as a non-responder if their week 24 (Visit 2) CAT score has

decreased by less than 2 units, has not changed, or has increased compared to the baseline CAT score. Baseline CAT score is as defined in Section 5.2.

 Ways of handling missing week 24 CAT score data are included in Section 7.1.1 as part of the estimands defined for this endpoint.

# **Secondary Endpoint**

#### **Multiple Lung Function Tests**

- If there are multiple spirometry tests recorded for a participant at <u>Visit 1</u>, the data from the latest test that
  is on or prior to the treatment start date will be considered in the planned data summaries and statistical
  analyses.
- If there are multiple spirometry tests recorded for a participant at <u>Visit 2</u>, the data from the latest test
  prior to study conclusion date will be considered for the planned data summaries and statistical
  analyses.

All lung function test data will be listed.

## Trough FEV<sub>1</sub>

For the spirometry assessment at Visit 1 and Visit 2, the following information is collected in the PFT dataset:

Q1: Please select the class of COPD maintenance treatment (Options: 9=ICS+LABA+LAMA; 10=LABA+LAMA; 12=ICS+LABA; 13=LABA; 14=LAMA)

**Q2:** (Goes with Q1) How long since the patient took their last dose of COPD maintenance treatment? (Options: **12**=0 to 4 hours; **13**=4 to 8 hours; **14**=8 to 12 hours; **15**=12 to 16 hours; **16**=16 to 24 hours; **17**=24 hours)

**Q3:** Please select the class of COPD maintenance treatment. If no additional maintenance to that provided in Q1 then please select "Not applicable". (Options: **9**=ICS+LABA+LAMA; **10**=LABA+LAMA; **12**=ICS+LABA; **13**=LABA; **14**=LAMA; "Not applicable")

**Q4:** (Goes with Q3) How long since the patient took their last dose of COPD maintenance treatment? Please select "Not applicable" if "Not applicable" selected in Q3. (Options: **12**=0 to 4 hours; **13**=4 to 8 hours; **14**=8 to 12 hours; **15**=12 to 16 hours; **16**=16 to 24 hours; **17**=24 hours; "Not applicable")

Trough FEV<sub>1</sub> will be defined as the FEV<sub>1</sub> value recorded while participants have withheld the COPD maintenance treatment.

- For COPD maintenance treatments taken <u>once-daily</u>, FEV<sub>1</sub> will be considered as Trough if the
  participant withheld the LABA and LAMA components of the maintenance treatment for at least 16 hours
  (category 16=16-24 hours or 17=24 hours selected in Q2 and Q4 (if applicable))
- For COPD maintenance treatments taken twice-daily, FEV<sub>1</sub> will be considered as Trough if the participant withheld the LABA and LAMA components of the maintenance treatment for at least 8 hours (category 14=8-12 hours, 15=12-16 hours, 16=16-24 hours or 17=24 hours selected in Q2 and Q4 (if applicable))

## Note:

- o If information is missing for some of the components of the maintenance COPD medication but available for the rest of the components, it will be assumed that the missing information is the same as the available information (e.g., if participant is on ICS + LABA + LAMA (MITT) and the LABA component was Trough but there is no information available for the LAMA component, then it will be assumed that LAMA component was also Trough. Similarly, if LABA component was recorded as non-Trough). Reminder: we do not consider the ICS as a monotherapy component for the definition of the Trough FEV1.
- o If information is completely missing for all components of the maintenance COPD medication, it will be assumed that the FEV<sub>1</sub> is not Trough.
- The maintenance COPD medication frequencies will be identified by linking the medication class selected at the PFT eCRF form with the medications listed in the Study Treatment eCRF form.

#### **Critical Errors**

- For the primary estimand of the secondary endpoint of critical errors (Section 7.2.3.4, Table 5), if
  participants modify their COPD maintenance therapy during the study the following scenarios are
  considered:
  - a) If the new therapy uses the same device(s) as the randomised COPD maintenance therapy, and error assessments are performed on these new device(s), this data will be used in the analysis.
  - b) If the new therapy uses different device(s) to the randomised COPD maintenance therapy, but they are device(s) that are assessed in the study (checklists available) and for which error assessments are performed, then this data will be set to missing.
  - c) If the new COPD maintenance therapy uses device(s) which are not being assessed in this study (no checklists available) then no error assessment is available at week 24 (Visit 2) and so this data is expected to be missing.
- For the supportive estimand of the secondary endpoint of critical errors, if participants modify their COPD maintenance therapy during the study the inhaler error data will be used regardless of whether the participant remained on the same device(s) after modifying the randomised treatment.
- According to the protocol, if participant is using more than one inhaler for the administration of the COPD maintenance therapy and inhaler error checklists are not available in the study for <u>all</u> the inhalers, then an inhaler error assessment should not be performed at Visit 2 by the participant. However, in the situation that an inhaler error assessment has been carried out for any of those inhalers for which a checklist is available, the data will not be used in the primary analyses (primary estimand) or the supportive analysis (supportive estimand) but they will be used in the exploratory analysis of the individual inhaler comparisons (Section 7.2.3.5.1).
- In the situation where a participant may miss a component of a device assessment and one or more of the other question responses (critical error) indicate an error was made, then the missing value has no additional impact on the response outcome as participant will be considered as having at least one critical error. In the situation where a participant may miss a component of a device assessment and all other responses to question indicate no error made, then the response to this endpoint (i.e., participant making at least one critical error) will be set to missing.

 More details around ways of handling missing week 24 CE data are included in Section 7.2.3 as part of the estimands defined for this endpoint.

## Other Endpoints

## Clinically Important Deterioration (CID)

CID is a composite outcome defined as any one of the following events:

- 1. 100 mL reduction from baseline in FEV<sub>1</sub> at 24 weeks. <u>Note:</u> Baseline <u>Trough</u> FEV<sub>1</sub> will be considered for this component.
- 2. An exacerbation (requiring treatment with antibiotics and/or systemic steroids or hospitalisation)
- 3. 2 units change (increase) from baseline in CAT score at 24 weeks

Note: Point 1 can only be considered for participants who are part of the  $FEV_1$  population (as defined in Section 4).

Ways of handling missing data in the analyses are included in Section 7.3.1 and Section 7.3.2 as part of the estimands defined for this endpoint.

For the listing of the CID data, the CID response flag will be defined as:

- If any of the three CID criteria defined above has been met, the participant will be considered as having experienced CID regardless of if the response to the other criteria is missing.
- If the response to any of the three CID criteria defined above is missing and the other criteria have not been met, then the CID response will be set to missing.

Note: The CID analyses incorporates multiple imputation for missing CAT score and missing Trough FEV<sub>1</sub> data as described in Section 7.3.1.4.

## **Time to First Moderate/Severe Exacerbation**

- Individual exacerbations are collected in the eCRF by the Investigator during the study.
  - COPD exacerbations will be classified as pre-randomised treatment, on-randomised treatment, post-randomised treatment, and on-study or post-study as described in Section 10.4.1.3. Also, exacerbation severity is defined in Section 10.6.1.
- The time to first exacerbation based only on on-randomised treatment data will be calculated as:

# [ First On-randomised Treatment Exacerbation Onset Date – Randomised Treatment Start Date ] + 1

Participants will be represented from the date of start of the randomised treatment to the start date of their first on-randomised treatment exacerbation or date of censoring. Participants that have not experienced an on-randomised treatment exacerbation are censored at the earliest of the randomised treatment stop date + 1 or the date of death.

• The time to first on-study exacerbation will be calculated as:

# [ First Exacerbation Onset Date – Randomisation Date ] + 1

Exacerbations reported during the on-study phase will be considered (see Section 10.4.1.3 for details of assigning study phase).

Participants will be represented from the day they were randomised in the study to the start date of their first exacerbation or date of censoring. Participants that have not experienced an on-study exacerbation are censored at the earliest of the study conclusion date or the date of death.

## **Annualised Rate of Moderate/Severe Exacerbations**

The annualized rate of on-randomised treatment exacerbations will be calculated as:

## [ Number of Exacerbations / Time on Randomised Treatment (in days) ] x 365.25

where:

| Number of Exacerbations: | Number of On-randomised Treatment Moderate/Severe<br>Exacerbations for each Participant |
|---|---|
| Time on Randomised Treatment: | [ earliest of (Randomised Treatment End Date + 1 or Date of Death or Study Conclusion Date) - Randomised Treatment Start Date ] +1 |

• The annualized rate of on-study exacerbations will be calculated as:

## [ Number of Exacerbations / Time on Study (in days) ] x 365.25

where:

| Number of Exacerbations: | Number of On-Study Moderate/Severe Exacerbations for each Participant |
|---|---|
| <u>Time on Study:</u> | [ earliest of (Study Conclusion Date or Study Withdrawal Date) - Randomisation Date ] +1 |

# **Exploratory Endpoints**

# Association of CE with CAT, moderate/ severe exacerbations, FEV1 and FVC

## • Association of CE with CAT score:

- A box-plot of the number of critical errors and the CAT score at week 24 will be populated. The number of errors (classified as: 0 errors; 1 error; ≥ 2 errors) will be presented on the x-axis and the week 24 CAT score (continuous) will be presented in the y-axis.
- A box-plot of the number of critical errors and the change from baseline in CAT score at week 24 will be populated. The number of errors (classified as: 0 errors; 1 error; ≥ 2 errors) will be presented on the x-axis and the change from baseline in CAT score at week 24 (continuous) will be presented in the y-axis.
- The number of critical errors (classified as: 0 errors; 1 error; ≥ 2 errors) and the CAT response at week 24 (classified as: Responders, Non-responders) will also be summarised in a frequency table.

#### Association of CE with FEV<sub>1</sub>:

A box-plot of the number of critical errors and the FEV<sub>1</sub> at week 24 will be populated. The number of

- errors (classified as: 0 errors; 1 error;  $\geq$  2 errors) will be presented on the x-axis and the week 24 FEV<sub>1</sub> (continuous) will be presented in the y-axis.
- A box-plot of the number of critical errors and the change from baseline in FEV₁ at week 24 will be
  populated. The number of errors (classified as: 0 errors; 1 error; ≥ 2 errors) will be presented on the
  x-axis and the change from baseline in FEV₁ at week 24 (continuous) will be presented in the y-axis.

## Association of CE with FVC:

- A box-plot of the number of critical errors and the FVC at week 24 will be populated. The number of
  errors (classified as: 0 errors; 1 error; ≥ 2 errors) will be presented on the x-axis and the week 24
  FVC (continuous) will be presented in the y-axis.
- O A box-plot of the number of critical errors and the change from baseline in FVC at week 24 will be populated. The number of errors (classified as: 0 errors; 1 error; ≥ 2 errors) will be presented on the x-axis and the change from baseline in FVC at week 24 (continuous) will be presented in the y-axis.

# • Association of CE with Moderate/Severe Exacerbations:

The number of critical errors (classified as: 0 errors; 1 error;  $\geq 2 \text{ errors}$ ) and the number of exacerbations (classified as: 0 exacerbations; 1 exacerbations; 2 exacerbations), will be summarised in a three-way frequency table. One frequency table for the on-randomised treatment moderate/severe exacerbations and one for the on-study moderate/severe exacerbations.

# Participant Treatment and Study Satisfaction Questionnaire

The Participant Treatment and Study Satisfaction Questionnaire include the following items:

| _ | CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are |
|---|---|
| • | protected by third party copyright laws and therefore have been excluded. |
| _ | |
| • | |

•

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

Data will be summarized and listed as described in Section 7.4.2.

# Health Related Quality of Life Questionnaire

The Health Related Quality of Life Questionnaire includes the following items:



Data will be summarised and listed as described in Section 7.4.3.

# 10.6.4. Safety

#### **Serious Adverse Events**

# **Serious Adverse Events of Special Interest**

SAESI have been defined as SAEs which have specified areas of interest for FF, VI or UMEC or the overall COPD population. The following table presents the SAESI groups. Groups which are not SMQs are made up of a selection of preferred terms (PTs) defined by GSK. The complete list, including the PTs which contribute to each of the groups will be provided by Global Clinical Safety and Pharmacovigilance (GCSP) using the MedDRA version current at the time of reporting. This will be finalized prior to unblinding.

| SAESI Group | SAESI Subgroup | Sub-SMQ |
|---|---|---|
| Cardiovascular effects | Cardiac arrhythmia Cardiac failure (SMQ) | Arrhythmia related investigations, signs and symptoms (SMQ) Bradyarrhythmia terms, nonspecific (SMQ) Conduction defects (SMQ) Disorders of sinus node function (SMQ) Cardiac arrhythmia terms, nonspecific (SMQ) Supraventricular tachyarrhythmias (SMQ) Tachyarrhythmia terms, nonspecific (SMQ) Ventricular tachyarrhythmias (SMQ) Ventricular tachyarrhythmias (SMQ) |
| | Ischaemic heart disease (SMQ) | |
| | Hypertension (SMQ) | |
| | Central nervous system haemorrhages and cerebrovascular conditions (SMQ) | |
| Decreased bone mineral density and associated fractures | | |
| Pneumonia | | Infective pneumonia SMQ (Narrow) |
| Lower Respiratory Tract Infection (LRTI) excluding pneumonia SMQ (Narrow) | | |

# For the planned summary of SAESI by class of medication:

- For the SAESI group of Pneumonia, events will be allocated to the treatment the participant was taking for the majority of the 28 days prior to the onset of the event. If the event occurred within 28 days of Randomisation, only the treatment taken post Randomisation is considered for the treatment allocation. For all other special interest groups, events are allocated to the treatment the participant was taking on the day of onset of the event.
- For SAESI group of Pneumonia, a participant will be considered at risk for a given treatment up until 28 days after the stop date of this treatment.

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e., as specified in the protocol) is defined as completion of the week 24 study visit (Visit 2). |
| | Participant treatment completion is defined as no premature discontinuation or modification of the randomised COPD maintenance treatment at any time prior to formal study completion. |
| | Withdrawn participants were not replaced in the study. |
| | ICH-required data from participants who were withdrawn from the study will be listed and all available planned data will be included in relevant summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |

Handling of missing data in the statistical analyses of the primary, secondary or other endpoints (i.e., *CID*), is described in Section 7 as part of the estimands framework. When multiple imputation is the suggested method for handling missing data, then the imputation will follow the steps described below.

| Element | Reporting Detail |
|---|---|
| Week 24<br>CAT | For the Primary Estimand and the Supportive Estimand II defined in Section 7.1.1.4 and Section 7.1.1.5.1, respectively, missing week 24 CAT score data will be imputed as described below: |
| | <ol> <li>In the original analysis dataset (Dataset A), a flag variable for each intercurrent event<br/>identified for the endpoint will be created, which will indicate the participants for which<br/>the intercurrent event has occurred.</li> </ol> |
| | <ol> <li>If a participant has reported at least one intercurrent event for which a "composite"<br/>strategy is suggested, the continuous endpoint data (if available) for that participant<br/>will be set to missing. All participants remain in one dataset which will be used for the<br/>imputation.</li> </ol> |
| | 3. First step of the imputation will be to run an imputation model (parameter-estimation model) to get pseudo-independent samples from the joint posterior distribution for the linear predictor parameters ("betas" associated with treatment, baseline CAT score (continuous), number of exacerbations in the prior year (categorical), prior medication |
use strata (categorical) and country (categorical)) and the covariance parameters.

- 4. Next step is to impute the missing endpoint data (as continuous data) by constructing endpoint estimates from the samples. This will be done assuming that the data is missing-at-random (MAR) i.e., based on the randomised treatment arm characteristics. A sufficient number of *m* samples (imputations) will be used to ensure that the final estimates are consistent and independent of any seeds used in the sampling process. Note that the participants with an intercurrent event for which a composite strategy is planned, will technically also have their "missing" continuous data imputed but this will be ignored. Also, note that participants with missing baseline CAT score (or any other missing covariates) will not be included in the analysis as they will not have a change from baseline.
- 5. There will be *m* imputed sets of data for analysis.
- 6. For each set of data, a binary response variable indicating responders and non-responders based on the change from baseline CAT score at week 24 (Visit 2) will be created for each participant. Note that the imputed continuous data for those participants flagged as having a composite intercurrent event should be set back to missing and the response status defined as "non-response" by definition (composite strategy).
- 7. A univariate logistic regression analysis will be performed for each set of data as described in Section 7.1.1.5.1.
- 8. The "m" results from the analyses of each set of data are combined using Rubin's formulae [Rubin, 1987]. (Note: model estimates should be combined on the model scale rather than the exponentiated [odds ratio] scale and then turned into an odds ratio by exponentiating).

**Note:** This approach will also be used for the imputation of missing CAT score data for the analysis of 2 Units Change (Increase) from Baseline in CAT score at 24 weeks (CID analysis of components, Section 7.3.2.2), adjusting for the covariates specified for this analysis (i.e., baseline CAT, prior medication use strata and country) and for the imputation of missing Trough FEV<sub>1</sub> data for the analysis of 100mL reduction in Trough FEV<sub>1</sub> at 24 weeks (analysis of CID components, Section 7.3.2.1), adjusting for the covariates specified for these analyses (i.e., baseline Trough FEV<sub>1</sub>, prior medication use strata and country.

For the Supportive Estimand III (Hypothetical) defined in Section 7.1.1.5.1, week 24 CAT score data will be imputed as described below:

- 1. In the original analysis dataset (Dataset A), a flag variable for each intercurrent event identified for the endpoint will be created, which will indicate the participants for which the intercurrent event has occurred.
- 2. For participants who have reported any of the intercurrent events identified for the endpoint, their response (if available) after the occurrence of the event (i.e., week 24 (Visit 2) CAT score) will be set to missing (Dataset B). All missing week 24 (Visit 2) CAT score values (those originally missing and those set to missing) will be imputed. Dataset B will be used for the imputation.
- 3. First step of the imputation will be to run an imputation model (parameter-estimation model) to get pseudo-independent samples from the joint posterior distribution for the linear predictor parameters ("betas" associated with treatment, baseline CAT score

- (continuous), number of exacerbations in the prior year (categorical), prior medication use strata (categorical) and country (categorical)) and the covariance parameters.
- 4. Next step is to impute the missing endpoint data (as continuous data) by constructing endpoint estimates from the samples. This will be done assuming that the data is missing-at-random (MAR) i.e. based on the randomised treatment arm characteristics. A sufficient number of *m* samples (imputations) will be used to ensure that the final estimates are consistent and independent of any seeds used in the sampling process.
- 5. There will be *m* imputed sets of data for analysis.
- 6. For each set of data for analysis, a binary response variable indicating the responders and non-responders based on the change from baseline CAT score at week 24 (Visit 2) will be created for each participant.
- 7. A univariate logistic regression analysis will be performed for each "new" analysis dataset as described in RAP Section 7.1.1.5.1.
- 8. The "m" results from the analyses of each dataset are combined using Rubin's formulae [Rubin, 1987]. (Note: model estimates should be combined on the model scale rather than the exponentiated [odds ratio] scale and then turned into an odds ratio by exponentiating).

#### Week 24 FEV<sub>1</sub>/ Trough FEV<sub>1</sub>

For the estimands defined in Sections 7.2.1 (FEV<sub>1</sub> analysis) and Section 7.2.2 (Trough FEV<sub>1</sub> analysis), missing week 24 FEV<sub>1</sub>/Trough FEV<sub>1</sub> data will be imputed as described below:

- 1. In the original analysis dataset (Dataset A), a flag variable for each intercurrent event identified for the endpoint will be created, which will indicate the participants for which the intercurrent event has occurred
- 2. Note that for the intercurrent events defined for these endpoints, no composite strategy is planned so Dataset A will be used as it is for the imputation.
- 3. First step of the imputation will be to run an imputation model (parameter-estimation model) to get pseudo-independent samples from the joint posterior distribution for the linear predictor parameters ("betas" associated with treatment, baseline FEV<sub>1</sub>/Trough FEV<sub>1</sub> score (continuous), prior medication use strata (categorical), country (categorical) and timing of spirometry (categorical only for the FEV<sub>1</sub> analysis)) and the covariance parameters.
- 4. Next step is to impute the missing endpoint data (as continuous data) by constructing endpoint estimates from the samples. This will be done assuming that the data is missing-at-random (MAR) i.e. based on the randomised treatment arm characteristics. A sufficient number of m samples (imputations) will be used to ensure that the final estimates are consistent and independent of any seeds used in the sampling process.
  - Note that participants with missing  $FEV_1/Trough\ FEV_1$  at Visit 1 (or any other missing covariates) will not be included in the analysis as they will not have a change from baseline.
- 5. There will be *m* imputed sets of data for analysis.
- 6. For each set of data, a univariate ANCOVA analysis will be performed for each set of

data as described in Section 7.2.1.5.1 (FEV $_1$  analysis) and Section 7.2.2.5.1 (Trough FEV $_1$  analysis).

7. The "m" results from the analyses of each set of data are combined using Rubin's formulae [Rubin, 1987].

#### CID

For the estimand defined in Section 7.3.1.4, missing week 24 CAT score data and/or missing week 24 Trough FEV<sub>1</sub> data will be imputed as described below:

- 1. In the original analysis dataset (Dataset A), a flag variable for each intercurrent event identified for the endpoint will be created, which will indicate the participants for which the intercurrent event has occurred.
- 2. If a participant has reported at least one intercurrent event for which a "composite" strategy is suggested, the continuous week 24 Trough FEV<sub>1</sub> data and the CAT score data for that participant (if available) will be set to missing. All participants remain in the one dataset which will be used for the imputation.
- 3. For each of the following components of the CID endpoint: a) CAT score and b) Trough FEV<sub>1</sub>, first step of the imputation will be to run an imputation model (parameter-estimation model) to get pseudo-independent samples from the joint posterior distribution for the linear predictor parameters ("betas" associated with treatment, baseline Trough FEV<sub>1</sub> (continuous), baseline CAT score (continuous), number of exacerbations in the prior year (categorical), prior medication use strata (categorical) and country (categorical)) and the covariance parameters. Note: Missing exacerbation data will not be imputed.
- 4. For each of the components of the CID mentioned in the previous step (CAT score and Trough FEV<sub>1</sub>) next step is to impute the missing data (CAT score and Trough FEV<sub>1</sub> data) as continuous data by constructing endpoint estimates from the samples. This will be done assuming that the data is missing-at-random (MAR) i.e. based on the randomised treatment arm characteristics. A sufficient number of *m* samples (imputations) will be used to ensure that the final estimates are consistent and independent of any seeds used in the sampling process. Note that the participants with an intercurrent event for which a composite strategy is planned, will technically also have their "missing" continuous data imputed but this will be ignored. Also, note that participants with missing CAT score at Visit 1 or missing Trough FEV<sub>1</sub> data at Visit 1 (or any other missing covariates) will not be included in the analysis as they will not have a change from baseline.
- 5. There will be *m* imputed sets of data for analysis.
- 6. For each set of data, a binary response variable indicating participants who experience CID and those who do not (as defined in Section 10.6.3) will be created for each participant. Note that the imputed continuous data for those participants flagged as having a composite intercurrent event, should be set back to missing and the response status defined as "non-response" by definition (composite strategy).
- 7. A univariate logistic regression analysis will be performed for each set of data as described in Section 7.3.1.5.1.
- 8. The "m" results from the analyses of each set of data are combined using Rubin's formulae [Rubin, 1987]. (Note: model estimates should be combined on the model

| scale rather than the exponentiated [odds ratio] scale and then turned into an odds |
|---|
| ratio by exponentiating). |

## 10.7.2.1. Handling of Missing and Partial Dates

| Partial dates will be displayed as captured in participant listing displays. | Element | Reporting Detail |
|---|---|---|
| Treatment Stop Date randomised treatment discontinuation or randomised treatment modification) and has a missing or partial randomised treatment stop date, then the randomised treatment stop date will be imputed in the following way: If the date is completely missing, it will be imputed as the latest of Study Conclusion Date/ Visit 2 Date If partial date is available (only month and year available), then the day will be imputed as the earliest of [the Last Day of the Month or the Study Conclusion Date Visit 2 Date] If a partial date is available (only year available), then the day and month will be imputed as the earliest of [the Last Day of the Year or the Study Conclusion Date/ Visit 2 Date] If participant has discontinued from randomised treatment or modified randomised treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment stop date, then the randomised treatment stop date will be imputed in the following way: If the date is completely missing, it will be imputed as the Day Prior to the Start Date of the Modified Maintenance Treatment If a partial date is available (only month and year available), then the day will be imputed as the earliest of [the Last Day of the Month or the Day Prior to the Start Date of the Modified Maintenance Treatment] If a partial date is available (only year available), then the day and month will be imputed as the earliest of [the Last Day of the Year or the Day Prior to the Start Date of the Modified Maintenance Treatment] In the special situation where, a participant has discontinued from randomised treatment or modified randomised treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment start date will be imputed in the following way: If partial dates are available (only month and year available), and Visit 2 or Conclusion Date (if Visit 2 Date not available or Visit 2 Date = Conclusion Date) is in the same month, then the Modified Tre | General | Partial dates will be displayed as captured in participant listing displays. |
| treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment stop date, then the randomised treatment stop date will be imputed in the following way: If the date is completely missing, it will be imputed as the Day Prior to the Start Date of the Modified Maintenance Treatment If a partial date is available (only month and year available), then the day will be imputed as the earliest of [the Last Day of the Month or the Day Prior to the Start Date of the Modified Maintenance Treatment] If a partial date is available (only year available), then the day and month will be imputed as the earliest of [the Last Day of the Year or the Day Prior to the Start Date of the Modified Maintenance Treatment] In the special situation where, a participant has discontinued from randomised treatment or modified randomised treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment stop date, but the start date of the modified maintenance treatment is also missing or partial, then the randomised treatment stop date and the modified randomised treatment start date will be imputed in the following way: If partial dates are available (only month and year available), and Visit 2 or Conclusion Date (if Visit 2 Date not available or Visit 2 Date = Conclusion Date) is in the same month, then the Modified Treatment Start Date will be imputed as the | Treatment | randomised treatment discontinuation or randomised treatment modification) and has a missing or partial randomised treatment stop date, then the randomised treatment stop date will be imputed in the following way: O If the date is completely missing, it will be imputed as the latest of Study Conclusion Date/ Visit 2 Date O If partial date is available (only month and year available), then the day will be imputed as the earliest of [the Last Day of the Month or the Study Conclusion Date Visit 2 Date] O If a partial date is available (only year available), then the day and month will be imputed as the earliest of [the Last Day of the Year or the Study Conclusion Date/ |
| treatment or modified randomised treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment stop date, but the start date of the modified maintenance treatment is also missing or partial, then the randomised treatment stop date and the modified randomised treatment start date will be imputed in the following way: o If partial dates are available (only month and year available), and Visit 2 or Conclusion Date (if Visit 2 Date not available or Visit 2 Date = Conclusion Date) is in the same month, then the Modified Treatment Start Date will be imputed as the | | treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment stop date, then the randomised treatment stop date will be imputed in the following way: o If the date is completely missing, it will be imputed as the Day Prior to the Start Date of the Modified Maintenance Treatment o If a partial date is available (only month and year available), then the day will be imputed as the earliest of [the Last Day of the Month or the Day Prior to the Start Date of the Modified Maintenance Treatment] o If a partial date is available (only year available), then the day and month will be imputed as the earliest of [the Last Day of the Year or the Day Prior to the Start |
| the Day Prior to the Imputed Modified Treatment Stop Date. E.g., Date Original Date Imputed Date | | treatment or modified randomised treatment during the study or discontinued from study (Early Withdrawal) and has a missing or partial randomised treatment stop date, but the start date of the modified maintenance treatment is also missing or partial, then the randomised treatment stop date and the modified randomised treatment start date will be imputed in the following way: o If partial dates are available (only month and year available), and Visit 2 or Conclusion Date (if Visit 2 Date not available or Visit 2 Date = Conclusion Date) is in the same month, then the Modified Treatment Start Date will be imputed as the Day Prior to Visit 2/ Conclusion Date and the Randomised Treatment Stop Date as the Day Prior to the Imputed Modified Treatment Stop Date. E.g., |
| Randomised Treatment Stop DateApr-2019 22-Apr-2019 | | <u> </u> |
| Modified Treatment Start DateApr-2019 23-Apr-2019 | | |

| Element | Reportir | ng Detail | | |
|---|---|---|---|---|
| | | Visit 2 Date | 24-Apr-2019 | N/A |
| | | For the scenario above, same rule will app missing but the other is partial or if both da | | |
| | o If partial dates are available (only month and year available), and Visit 2 or Conclusion Date (if Visit 2 date not available or Visit 2 Date = Conclusion Date) not in the same month, then the Modified Treatment Start Date will be imputed the Last Day of the Month (of the partial date) and the Randomised Treatment Start Date as the Day Prior to the Imputed Modified Treatment Stop Date. E.g., | | | |
| | | Date | Original Date | Imputed Date |
| | | Randomised Treatment Stop Date | Apr-2019 | 29-Apr-2019 |
| | | Modified Treatment Start Date | Apr-2019 | 30-Apr-2019 |
| | | Visit 2 Date | 10-May-2019 | N/A |
| | | For the scenario above, if the Randomised Treatment Stop Date is partial and the Modified Treatment Start Date dates is completely missing, then the Randomised Treatment Stop Date will be imputed as the last day of the month (of the partial date) and the Modified Treatment Start Date as the Day After the Imputed Randomised Treatment Stop Date. | | |
| Adverse<br>Events/ | | <ul> <li>The eCRF does not allow for the possibility of partial dates to be recorded for AE/SAE<br/>start and end dates.</li> </ul> | | |
| Serious<br>Adverse<br>Events | | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. | | |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> | | | |

# 10.8. Appendix 8: Abbreviations & Trade Marks

### 10.8.1. Abbreviations

| Abbreviation | Description |
|------------------|------------------------------------------------|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CAT | COPD Assessment Test |
| CDISC | Clinical Data Interchange Standards Consortium |
| CE | Critical Error |
| CI | Confidence Interval |
| CID | Clinically Important Deterioration |
| CIL | Clinical Investigation Lead |
| COPD | Chronic Obstructive Pulmonary Disease |
| CSR | Clinical Study Report |
| CV | Cardiovascular |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| DQL | Data Quality Lead |
| eCRF | Electronic Case Record Form |
| EHR | Electronic Health Record |
| EMA | European Medicines Agency |
| EW | Early Withdrawal |
| FDA | Food and Drug Administration |
| FEV <sub>1</sub> | Forced Expiratory Volume in 1 Second |
| FVC | Forced Vital Capacity |
| GOLD | Global Initiative on Obstructive Lung Disease |
| GSK | GlaxoSmithKline |
| HCP | Health Care Provider |
| HCRU | Healthcare Resource Utilisation |
| HRQoL | Health Related Quality of Life Questionnaire |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| IWRS | Interactive Web Response System |
| ITT | Intent-To-Treat |
| MAR | Missing at Random |
| MDI | Metered Dose Inhaler |
| MITT | Multiple Inhaler Triple Therapy |
| MM | Medical Monitor |
| OSL | Operational Study Lead |
| PDMP | Protocol Deviation Management Plan |
| PFT | Pulmonary Function Test |
| PP | Per Protocol |

| Abbreviation | Description |
|--------------|--------------------------------------------|
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RW | Real World |
| SAC | Statistical Analysis Complete |
| SERM | Safety Evaluation and Risk Management |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| VEO | Value Evidence and Outcomes |

## 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| CAT |
| DISKUS |
| ELLIPTA |
| RAMOS NG |
| RANDALL NG |
| TRELEGY |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| BREEZHALER |
| GENUAIR |
| HANDIHALER |
| SAS |
| TURBUHALER |

## 10.9. Appendix 9: List of Data Displays

### 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-----------------------|------------|
| Study Population | 1.1 to 1.n 1.1 to 1.n | |
| Effectiveness | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n N/A | |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | x+1 to y | |

### 10.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Effectiveness | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | - | SAFE_Tn | SAFE_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 10.9.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | ASE | Non-Standard | Summary of Subject Populations and Reasons for Screen Failure | | SAC |
| 1.2. | ITT | Non-Standard | Summary of Attendance at Each Visit by Visit Type | See IMPACT 1.02. For Visit 1, Visit type will be: 1) Patient usual care site; 2) Referral site; 3) Home visit. For Visit 2, Visit type will be the ones defined for Visit 1 with the addition of 4) Telephone Visit. Present EW visit separately using the Visit type categories defined for Visit 2. | SAC |
| 1.3. | FEV1 | Non-Standard | Summary of Attendance at Each Visit by Visit Type | As for Table 1.2. | SAC |
| 1.4. | CE | Non-Standard | Summary of Attendance at Each Visit by Visit Type | As for Table 1.2. | SAC |
| 1.5. | ITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC |
| 1.6. | FEV1 | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC |
| 1.7. | CE | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | ITT | ES1 | Summary of Study Status and Reasons for Study Withdrawal | | SAC |
| 1.9. | FEV1 | ES1 | Summary of Study Status and Reasons for Study Withdrawal | | SAC |
| 1.10. | CE | ES1 | Summary of Study Status and Reasons for Study Withdrawal | | SAC |
| 1.11. | ITT | Non-Standard | Summary of Prior Medication Use Strata | | SAC |
| 1.12. | ASE | Non-Standard | Summary of Number of Subjects by Country | Based on IDSL NS1 but display presented only by Country (not by Centre ID and Investigator ID). Only Total column is required. | SAC |
| 1.13. | ITT | NS1 | Summary of Number of Subjects by Country and Centre | | SAC |
| 1.14. | ASE | IE1 | Summary of Inclusion/Exclusion Criteria Deviations for Screen Failures | | SAC |
| 1.15. | ITT | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC |
| Protoc | ol Deviation | | | | |
| 1.16. | ITT | DV1 | Summary of Important Protocol Deviations | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.17. | ASE | DM11 | Summary of Age Ranges | As per IDSL DM11 but also see<br>Section 10.6.2. | SAC |
| 1.18. | ITT | DM1 | Summary of Demographic Characteristics | As per IDSL DM1 but also see<br>Section 10.6.2. | SAC |
| 1.19. | FEV1 | DM1 | Summary of Demographic Characteristics | As per IDSL DM1 but also see<br>Section 10.6.2. | SAC |
| 1.20. | CE | DM1 | Summary of Demographic Characteristics | As per IDSL DM1 but also see<br>Section 10.6.2. | SAC |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.21. | ITT | DM1 | Summary of Demographic Characteristics by Country | | SAC |
| 1.22. | ITT | DM1 | Summary of Demographic Characteristics by Prior Medication Use Strata | | SAC |
| 1.23. | ITT | DM5 | Summary of Race and Racial Combinations | As per IDSL DM5 but also see<br>Section 10.6.2. | SAC |
| Medica | I Conditions | | | | |
| 1.24. | ITT | MH4 | Summary of Current Medical Conditions | | SAC |
| 1.25. | ITT | MH4 | Summary of Past Medical Conditions | | SAC |
| 1.26. | ITT | Non-Standard | Summary of Cardiovascular Risk Factors | | SAC |
| 1.27. | ITT | FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| Diseas | e Characteristic | cs | | | |
| 1.28. | ITT | Non-Standard | Summary of COPD Duration at Screening | | SAC |
| 1.29. | ITT | Non-Standard | Summary of COPD Exacerbation History at Screening | | SAC |
| 1.30. | FEV1 | Non-Standard | Summary of Lung Function at Screening | Table will include all available Screening data regardless of visit type (e.g., domiciliary visit etc). It will also include historical CAT score data (more than 14 days prior to V1 - not flagged as baseline). | SAC |
| 1.31. | FEV1 | Non-Standard | Summary of Reversibility and GOLD Grade (1-4) at Screening | See Section 10.6.2. | SAC |
| 1.32. | FEV1 | Non-Standard | Summary of PIFR (L/min) at Screening | | SAC |
| 1.33. | ITT | Non-Standard | Summary of CAT Score and CAT Category at Screening | CAT categories: CAT < 10 and CAT ≥ 10. | SAC |
| 1.34. | ITT | Non-Standard | Summary of Historical Eosinophils Data | See Section 10.6.2. | SAC |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | • |
| 1.35. | ITT | Non-Standard | Summary of Pre-randomised Treatment Respiratory Concomitant Medications Excluding those Taken for an Exacerbation | Non-Standard but based on IDSL<br>CM1. RMC classification to be<br>used. | SAC |
| 1.36. | ITT | Non-Standard | Summary of On-randomised Treatment Respiratory<br>Concomitant Medications Excluding those Taken for an<br>Exacerbation | Non-Standard but based on IDSL<br>CM1. RMC classification to be<br>used. Randomised COPD<br>Maintenance Therapy will not be<br>included in this summary. | SAC |
| 1.37. | ITT | Non-Standard | Summary of Post-randomised Treatment Respiratory Concomitant Medication Excluding those Taken for an Exacerbation | Non-Standard but based on IDSL<br>CM1. RMC classification to be<br>used. | SAC |
| 1.38. | ITT | Non-Standard | Summary of Pre-randomised Treatment COPD Concomitant Medications Taken for an Exacerbation | Non-Standard but based on IDSL<br>CM1. RMC classification to be<br>used. | SAC |
| 1.39. | ITT | Non-Standard | Summary of On-randomised Treatment COPD Concomitant Medications Taken for an Exacerbation | Non-Standard but based on IDSL CM1. RMC classification to be used. | SAC |
| 1.40. | ITT | Non-Standard | Summary of Post-randomised Treatment COPD Concomitant Medications Taken for an Exacerbation | Non-Standard but based on IDSL CM1. RMC classification to be used. | SAC |
| 1.41. | ITT | Non-Standard | Summary of Respiratory Concomitant Medication Combinations Taken at Screening Excluding Those Taken for an Exacerbation | Non-Standard but based on IDSL<br>CM1. RMC classification to be<br>used. See IMPACT Table 1.67. | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.42. | ITT | Non-Standard | Summary of Respiratory Concomitant Medication Taken at Treatment Discontinuation Excluding Those Taken for an Exacerbation | Non-Standard but based on IDSL<br>CM1. RMC classification to be<br>used. See IMPACT Table 1.70. | SAC |
| Treatm | ent Exposure | | | | |
| 1.43. | ITT | Non-Standard | Summary of Treatment Exposure | Exposure to Randomised Treatment. Also present the total time in study post-randomised treatment and the total time spent on-study. See 207609 Table 3.1. | SAC |
| 1.44. | ITT | Non-Standard | Summary of Unique Treatment Paths | See study HZC115151, Table 1.34 (only bottom segment is required). | SAC |
| Intercu | rrent Events | | | | |
| 1.45. | ITT | Non-Standard | Summary of Intercurrent Events | | SAC |
| 1.46. | FEV1 | Non-Standard | Summary of Intercurrent Events | | SAC |
| 1.47. | CE | Non-Standard | Summary of Intercurrent Events | | SAC |

# 10.9.5. Study Population Figures

| Study P | Study Population Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.1. | ITT | Non-Standard | Kaplan-Meier Plot of Time to Premature Discontinuation of Study Treatment | | SAC |
| 1.2. | ITT | Non-Standard | Kaplan-Meier Plot of Time to Study Withdrawal | | SAC |

### 10.9.6. Effectiveness Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | / Endpoint | | | | |
| 2.1. | ITT | Non-Standard | Summary of CAT Score | Summary at each visit (Baseline CAT, Week 24 and Change from Baseline – separate out EW visit). | SAC |
| 2.2. | ITT | Non-Standard | Summary and Analysis of the Percentage of Responders<br>According to the CAT Score at Week 24 (Primary Estimand -<br>Treatment Policy x Composite) | Include Footnote: "Note: A Treatment policy strategy was used for the intercurrent event of Randomised Treatment Discontinuation. For the intercurrent events of Randomised Treatment Modification, change of Pulmonary Rehabilitation status and start of Oxygen Therapy, a Composite strategy was used." | SAC |

| Efficacy | /: Tables | T | | I | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | ITT | Non-Standard | Summary and Analysis of the Percentage of Responders<br>According to the CAT Score at Week 24 (Supportive Estimand I-<br>Treatment Policy x Composite) | Include Footnote: "Note: A Treatment policy strategy was used for the intercurrent event of Randomised Treatment Discontinuation, Randomised Treatment Modification, change of Pulmonary Rehabilitation status and start of Oxygen Therapy. Subjects who prematurely discontinue from study and subjects with missing Visit 2 (Week 24) CAT score (for other reason) are considered as non-responders". | SAC |
| 2.4. | ITΤ | Non-Standard | Summary and Analysis of the Percentage of Responders According to the CAT Score at Week 24 (Supportive Estimand II– Treatment Policy x Composite) | Include Footnote: "Note: A Treatment policy strategy was used for the intercurrent events of Randomised Treatment Discontinuation, change of Pulmonary Rehabilitation status and start of Oxygen Therapy. For the intercurrent event of Randomised Treatment Modification, a Composite strategy was used." | SAC |

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.5. | ITT | Non-Standard | Summary and Analysis of the Percentage of Responders<br>According to the CAT Score at Week 24 (Supportive Estimand<br>III– Hypothetical) | Include Footnote: "Note: A Hypothetical strategy was used for the intercurrent events of Randomised Treatment Discontinuation, Randomised Treatment Modification, change of Pulmonary Rehabilitation status and start of Oxygen Therapy.". | SAC |
| 2.6. | ITT | Non-Standard | P-values for Interactions of Treatment with Covariates for<br>Analysis of the Percentage of Responders According to the CAT<br>Score at Week 24 (Primary Estimand - Treatment Policy x<br>Composite) | The p-value for each interaction test will be presented. If any interaction p-value is less than 0.10 further investigations will be carried out, for example running the analysis by each category of the subgroup. Any output from interaction investigation will also be presented in additional displays. | SAC |
| Second | ary Endpoints | | | | |
| 2.7. | FEV1 | Non-Standard | Summary of FEV1 | Summary at each visit (Baseline FEV1, Week 24 and Change from Baseline – separate out EW visit). | SAC |
| 2.8. | FEV1 | Non-Standard | Summary of Trough FEV1 | Summary at each visit (Baseline<br>Trough FEV1, Week 24 and<br>Change from Baseline – separate<br>out EW visit). | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.9. | FEV1 | Non-Standard | Analysis of Change from Baseline in FEV1 at Week 24 (Primary Estimand – Treatment Policy) | Include Footnote: "Note: A Treatment Policy strategy was used for the intercurrent events of Randomised Treatment Discontinuation, Randomised Treatment Modification, change of Pulmonary Rehabilitation status and start of Oxygen Therapy." | SAC |
| 2.10. | FEV1 | Non-Standard | Analysis of Change from Baseline in Trough FEV1 at Week 24 (Primary Estimand – Treatment Policy) | Include Footnote: "Note: A Treatment Policy strategy was used for the intercurrent events of Randomised Treatment Discontinuation, Randomised Treatment Modification, change of Pulmonary Rehabilitation status and start of Oxygen Therapy." | SAC |
| 2.11. | CE | Non-Standard | Summary of Critical and Overall Errors | Each inhaler presented on different page. Frequency for each error type to be presented for each inhaler. Flag with "[1]" the error types which are considered as critical errors and include relevant footnote. Include footnote: "All inhalers apart from the Ellipta inhaler are used in combination with at least one other inhaler by the subjects." | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | CE | Non-Standard | Analysis of the Percentage of Subjects Making at Least One<br>Critical Error at Week 24 (Primary Estimand – Hypothetical) | Include Footnote: "Note: A Hypothetical strategy was used for the intercurrent event of Randomised Treatment Modification.". | SAC |
| 2.13. | CE | Non-Standard | Analysis of the Percentage of Subjects Making at Least One<br>Critical Error at Week 24 (Supportive Estimand – Treatment<br>Policy) | Include Footnote: "Note: A Treatment Policy strategy was used for the intercurrent event of Randomised Treatment Modification.". | SAC |
| 2.14. | ITT | Non-Standard | Analysis of the Percentage of Subjects Making at Least One<br>Critical Error at Week 24 Ellipta vs Comparator Device<br>(Exploratory Estimand – Treatment Policy) | Exploratory analysis to be performed if at least 100 subjects/arm perform an inhaler assessment. Comparison of inhalers: Ellipta vs Diskus; Ellipta vs Breezhaler; Ellipta vs Handihaler; Ellipta vs MDI; Ellipta vs Turbuhaler; Ellipta vs Genuair to be presented in each page. | SAC |
| Other E | ndpoints | | | · | |

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.15. | FEV1 | Non-Standard | Summary and Analysis of the Percentage of Subjects Who Experience Clinically Important Deterioration (Primary Estimand – Treatment Policy x Composite) | Include Footnote: "Note: A Treatment Policy strategy was used for the intercurrent events of Randomised Treatment Discontinuation, Randomised Treatment Modification and change of Pulmonary Rehabilitation status. For the intercurrent event of start of Oxygen Therapy, a Composite strategy was used." | SAC |
| 2.16. | FEV1 | Non-Standard | Summary and Analysis of the Percentage of Subjects Who Experience Clinically Important Deterioration (Sensitivity Analysis – Treatment Policy x Composite Estimand) | Same estimand as in Table 2.15, excluding the number of exacerbations in the prior year from the list of covariates in the model. | SAC |
| 2.17. | FEV1 | Non-Standard | Summary and Analysis of the Percentage of Subjects Who Experience a 100 mL Reduction from Baseline in Trough FEV1 at 24 Weeks (Primary Estimand – Treatment Policy x Composite) | Include Footnote: "Note: A Treatment Policy strategy was used for the intercurrent events of Randomised Treatment Discontinuation, Randomised Treatment Modification and change of Pulmonary Rehabilitation status. For the intercurrent event of start of Oxygen Therapy, a Composite strategy was used." | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18. | FEV1 | Non-Standard | Summary and Analysis of the Percentage of Subjects Who Experience a 2-unit Change (Increase) from Baseline in CAT Score at 24 Weeks (Primary Estimand – Treatment Policy x Composite) | Include Footnote: "Note: A Treatment Policy strategy was used for the intercurrent events of Randomised Treatment Discontinuation, Randomised Treatment Modification and change of Pulmonary Rehabilitation status. For the intercurrent event of start of Oxygen Therapy, a Composite strategy was used." | SAC |
| 2.19. | ITT | Non-Standard | Summary of On-randomised Treatment Moderate/Severe COPD Exacerbations | | SAC |
| 2.20. | ITT | Non-Standard | Summary of On-Study Moderate/Severe COPD Exacerbations | | SAC |
| 2.21. | ITT | Non-Standard | Summary of Annualised Rate of On-Study Moderate/Severe Exacerbations | | SAC |
| 2.22. | ITT | Non-Standard | Kaplan Meir Estimates of Time to First On-randomised<br>Treatment Moderate/Severe COPD Exacerbations | Just at Day 169. | SAC |
| 2.23. | ITT | Non-Standard | Kaplan Meir Estimates of Time to First On-Study<br>Moderate/Severe COPD Exacerbations | Just at Day 169. | SAC |
| 2.24. | ITT | Non-Standard | Summary of Unscheduled COPD Related Healthcare Contacts | | SAC |
| Explora | tory Endpoints | S | | | |
| 2.25. | CE | Non-Standard | Association of Number of Critical Errors and CAT Response at Week 24 | Frequency table. Categories as described in Section 10.6.3. | SAC |
| 2.26. | CE | Non-Standard | Association of Number of Critical Errors and On-randomised<br>Treatment Moderate/Severe Exacerbations | A 3-way frequency table. Categories as described in Section 10.6.3. | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27. | CE | Non-Standard | Association of Number of Critical Errors and On-Study<br>Moderate/Severe Exacerbations | A 3-way frequency table. Categories as described in Section 10.6.3. | SAC |
| 2.28. | ITT | Non-Standard | Summary of Subject Treatment and Study Satisfaction Questionnaire Responses at Week 24/ EW Visit | | SAC |
| 2.29. | ITT | Non-Standard | Summary of Health Related Quality of Life Questionnaire Responses | Summary at each Visit. | SAC |

# 10.9.7. Effectiveness Figures

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | y Endpoint | | | | <u> </u> |
| 2.1. | ITT | Non-Standard | Box-plot of Change from baseline in CAT Score at Week 24 | See Section 10.6.3. | SAC |
| Other E | Endpoints | | | | |
| 2.2. | ITT | Non-Standard | Kaplan Meir Plot for Time to First On-randomised Treatment Moderate/Severe Exacerbation | | SAC |
| 2.3. | ITT | Non-Standard | Kaplan Meir Plot for Time to On-Study First Moderate/Severe Exacerbation | | SAC |
| Explora | atory Endpoints | S | | | |
| 2.4. | CE | Non-Standard | Box-plot of Association of Critical Errors with CAT Score at Week 24 | See Section 10.6.3. | SAC |
| 2.5. | CE | Non-Standard | Box-plot of Association of Critical Errors with Change from Baseline in CAT Score at Week 24 | See Section 10.6.3. | SAC |
| 2.6. | CE | Non-Standard | Box-plot of Association of Critical Errors with FEV1 at Week 24 | See Section 10.6.3. | SAC |
| 2.7. | CE | Non-Standard | Box-plot of Association of Critical Errors with Change from Baseline in FEV1 at Week 24 | See Section 10.6.3. | SAC |
| 2.8. | CE | Non-Standard | Box-plot of Association of Critical Errors with FVC at Week 24 | See Section 10.6.3. | SAC |
| 2.9. | CE | Non-Standard | Box-plot of Association of Critical Errors with Change from Baseline in FVC at Week 24 | See Section 10.6.3. | SAC |

## 10.9.8. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | ITT | Non-Standard | Summary of Adverse Events Overview | byval: On-randomised Treatment, Post-randomised Treatment. Include Footnote: "Note: Only treatment related AEs and AEs that lead to withdrawal from study treatment and Serious AEs are collected and | SAC |
| 3.2. | ITT | AE1 | Summary of Pre-randomised Treatment Adverse Events by | summarised.". Same comments as for 3.1. Based on IDSL AE1 presenting also | SAC |
| J.Z. | | ALI | System Organ Class and Preferred Term | rates. Same comments as for 3.1. | UNO . |
| 3.3. | ITT | AE1 | Summary of On-randomised Treatment Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.4. | ITT | AE1 | Summary of Post-randomised Treatment Adverse Events by<br>System Organ Class and Preferred Term | Same comments as for 3.1. Based on IDSL AE1 presenting also rates. | SAC |
| 3.5. | ITT | AE1 | Summary of On-Study Adverse Events by System Organ Class and Preferred term | Same comments as for 3.1. Based on IDSL AE1 presenting also rates. | SAC |
| 3.6. | ITT | AE1 | Summary of On-randomised Treatment Drug-related Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.7. | ITT | AE1 | Summary of Post-randomised Treatment Drug-related Adverse<br>Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.8. | ITT | AE1 | Summary of On-randomised Treatment Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.9. | ITT | AE15 | Summary of Common (>=1% in Either Treatment Group) On-<br>randomised Treatment Non-serious Adverse Events by System<br>Organ Class and Preferred Term (Number of Subjects and<br>Occurrences) | Include Footnote: "Note: Only treatment related AEs and AEs that lead to withdrawal from study treatment are summarised." | SAC |
| Serious | and Other Sig | nificant Adverse l | Events | , , | |
| 3.10. | ITT | AE16 | Summary of On-randomised Treatment Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.11. | ASE | AE1 | Summary of Pre-randomised Treatment Serious Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.12. | ITT | AE1 | Summary of Pre-randomised Treatment Serious Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.13. | ITT | AE1 | Summary of On-randomised Treatment Serious Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.14. | ITT | AE1 | Summary of Post-randomised Treatment Serious Adverse<br>Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.15. | ITT | AE1 | Summary of On-Study Serious Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.16. | ITT | AE1 | Summary of On-randomised Treatment Serious Adverse Events<br>Leading to Permanent Discontinuation of Study Treatment or<br>Withdrawal from Study by System Organ Class and Preferred<br>Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.17. | ITT | AE1 | Summary of On-randomised Treatment Fatal Serious Adverse<br>Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.18. | ITT | AE1 | Summary of Post-randomised Treatment Fatal Serious Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.19. | ITT | Non-Standard | Summary of On-Study Fatal Serious Adverse Events by Class of Medication | | SAC |
| 3.20. | ITT | AE1 | Summary of Pre-randomised Treatment Serious Adverse Events<br>Leading to Withdrawal from Study by System Organ Class and<br>Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.21. | ITT | AE1 | Summary of On-randomised Treatment Drug-Related Serious Adverse Events by System Organ Class and Preferred Term | Based on IDSL AE1 presenting also rates. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.22. | ITT | AE1 | Summary of On-randomised Treatment Drug-Related Fatal<br>Serious Adverse Events by System Organ Class and Preferred<br>Term | Based on IDSL AE1 presenting also rates. | SAC |
| 3.23. | ITT | AE3 | Summary of Common (>=1% in Either Treatment Group) On-<br>randomised Treatment Serious Adverse Events by Preferred<br>Term | Present by PT (not SOC). | SAC |
| 3.24. | ITT | Non-Standard | Summary of On-randomised Treatment Serious Adverse Events of Special Interest | Based on IDSL AE1 but present by<br>Special Interest (SI) Group, SI<br>Subgroup, Sub-SMQ and PT. Also,<br>present rates. | SAC |
| 3.25. | ITT | Non-Standard | Summary of Post-randomised Treatment Serious Adverse<br>Events of Special Interest | Based on IDSL AE1 but present by<br>Special Interest (SI) Group, SI<br>Subgroup, Sub-SMQ and PT. Also,<br>present rates. | SAC |
| 3.26. | ITT | Non-Standard | Summary of On-Study Serious Adverse Events of Special Interest by Class of Medication | | SAC |

# 10.9.9. ICH Listings

All ICH listings will be presented by Country, unless otherwise specified.

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | ASE | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | ITT | TA1 | Listing of Randomised and Actual Treatments | | SAC |
| 3. | ITT | TA1 | Listing of Randomised and Actual Prior Medication Use Strata | | SAC |
| 4. | ITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 5. | ITT | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| Protoc | ol Deviations | | | | |
| 6. | ITT | DV2 | Listing of Important Protocol Deviations | | SAC |
| 7. | ASE | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations for Screen Failures | | SAC |
| 8. | ITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 9. | ITT | DM2 | Listing of Demographic Characteristics | | SAC |
| 10. | ITT | DM9 | Listing of Race | | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | ITT | Non-Standard | Listing of Respiratory Concomitant Medications | Including flag to indicate those taken for an exacerbation (COPD). | SAC |
| Treatm | ent Exposure | | | | |
| 12. | ITT | Non-Standard | Listing of Exposure Data | | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 13. | ASE | AE8 | Listing of All Adverse Events | Include Footnote: "Note: Only treatment related AEs and AEs that lead to withdrawal from study treatment and Serious AEs are collected and listed." | SAC |
| 14. | ASE | AE7 | Listing of Subject Numbers for Individual Adverse Events | Footnote from Listing 13 is applicable to this display. Listing not presented by Country. | SAC |
| Serious | and Other Sig | nificant Adverse | Events | - | |
| 15. | ASE | AE8 | Listing of Fatal Serious Adverse Events | | SAC |
| 16. | ASE | AE8 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| 17. | ASE | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 18. | ASE | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| 19. | ITT | AE8 | Listing of Serious Adverse Events of Special Interest | | SAC |

## 10.9.10. Non-ICH Listings

All Non-ICH listings will be presented by Country, unless otherwise specified.

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study | Population | | | | |
| 20. | ITT | Non-Standard | Listing of Study Treatment Misallocations | Similar to IDSL TA1. | SAC |
| 21. | ITT | Non-Standard | Listing of Randomised Treatment and Randomised Treatment Modifications | | SAC |
| 22. | ITT | MH2 | Listing of Medical Conditions | | SAC |
| 23. | ITT | Non-Standard | Listing of Family History of Cardiovascular Risk Factors | | SAC |
| 24. | ITT | Non-Standard | Listing of COPD Exacerbation History | | SAC |
| 25. | ITT | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text for Non-Respiratory Medications | | SAC |
| 26. | ITT | Non-Standard | Listing of f Historical Eosinophils Data | | SAC |
| Effecti | veness | | | | |
| 27. | ITT | Non-Standard | Listing of CAT Scores | | SAC |
| 28. | FEV1 | Non-Standard | Listing of Lung Function Data | Listing will also include PIFR data. | SAC |
| 29. | ITT | Non-Standard | Listing of Inhaler Critical and Overall Errors | | SAC |
| 30. | FEV1 | Non-Standard | Listing of Clinically Important Deterioration Data | | SAC |
| 31. | ITT | Non-Standard | Listing of COPD Exacerbations | | SAC |
| 32. | ITT | Non-Standard | Listing of Participant Treatment and Study Satisfaction Questionnaire Responses | | SAC |

| Non-ICI | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 33. | ITT | Non-Standard | Listing of Health Related Quality of Life Questionnaire (HRQoL) Responses | | SAC |
| Safety | | | | | |
| 34. | 34. ITT Non-Standard SAE Terms of Special Interest Listing not presented by Country. | | | | |
| 35. | ITT | AE7 | Listing of Subject Numbers for On-randomised Treatment Serious Adverse Events of Special Interest | Listing not presented by Country. | SAC |

# 10.9.11. Patient Profile Listings

| Patient | Profile: Listing | js | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | Population | | | | |
| 36. | ITT | Non-Standard | Listing of Arrhythmias | Include information required by IDSL standards. | SAC |
| 37. | ITT | Non-Standard | Listing of Congestive Heart Failure | Include information required by IDSL standards. | SAC |
| 38. | ITT | Non-Standard | Listing of Cerebrovascular Events/ Stroke/ Transient Ischemic Attack | Include information required by IDSL standards. | SAC |
| 39. | ITT | Non-Standard | Listing of Deep Vein Thrombosis/ Pulmonary Embolism | Include information required by IDSL standards. | SAC |
| 40. | ITT | Non-Standard | Listing of Myocardial Infarction/ Unstable Angina | Include information required by IDSL standards. | SAC |
| 41. | ITT | Non-Standard | Listing of Peripheral Arterial Thromboembolism | Include information required by IDSL standards. | SAC |
| 42. | ITT | Non-Standard | Listing of Pulmonary Hypertension | Include information required by IDSL standards. | SAC |
| 43. | ITT | Non-Standard | Listing of Revascularisation | Include information required by IDSL standards. | SAC |
| 44. | ITT | Non-Standard | Listing of Valvulopathy | Include information required by IDSL standards. | SAC |

# 10.10. Appendix 10: Example Mock Shells for Data Displays

The data display shells are contained in separate documents and are available upon request.